CLINICAL TRIAL: NCT02833350
Title: A Two-Cohort Randomized Phase II, Double-Blind, Parallel Group Study in Patients With Active Rheumatoid Arthritis Evaluating the Efficacy and Safety of GDC-0853 Compared With Placebo and Adalimumab in Patients With an Inadequate Response to Previous Methotrexate Therapy (Cohort 1) and Compared With Placebo in Patients With an Inadequate Response or Intolerance to Previous TNF Therapy (Cohort 2)
Brief Title: Safety and Efficacy Study of GDC-0853 Compared With Placebo and Adalimumab in Participants With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA29350; 2016-000335-40 (EudraCT Number)
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fenebrutinib; Adalimumab; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- Cohort 1: GDC-0853 High Dose + Adalimumab Placebo (Experimental): Participants of Cohort 1 will receive GDC-0853 high dose, orally once daily along with placebo matched to adalimumab, subcutaneously every 2 weeks (Q2W) starting on Day 1 for 12 weeks. Participants will remain on a stable background therapy of MTX 15-25 milligrams per week (mg/week) (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week are allowed only if there is clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigator's discretion.
  Interventions: Drug: GDC-0853; Drug: Folic Acid; Drug: MTX; Drug: Placebo
- Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo (Experimental): Participants of Cohort 1 will receive GDC-0853 low dose, orally once daily along with placebo matched to adalimumab, subcutaneously Q2W starting on Day 1 for 12 weeks. Participants will remain on a stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week are allowed only if there is clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigator's discretion.
  Interventions: Drug: GDC-0853; Drug: Folic Acid; Drug: MTX; Drug: Placebo
- Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo (Experimental): Participants of Cohort 1 will receive GDC-0853 mid dose, orally twice daily along with placebo matched to adalimumab, subcutaneously Q2W starting on Day 1 for 12 weeks. Participants will remain on a stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week are allowed only if there is clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigator's discretion.
  Interventions: Drug: GDC-0853; Drug: Folic Acid; Drug: MTX; Drug: Placebo
- Cohort 1: GDC-0853 Placebo + Adalimumab (Active Comparator): Participants of Cohort 1 will receive placebo matched to GDC-0853, orally once daily along with adalimumab, subcutaneously Q2W starting on Day 1 for 12 weeks. Participants will remain on a stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week are allowed only if there is clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigator's discretion.
  Interventions: Drug: Adalimumab; Drug: Folic Acid; Drug: MTX; Drug: Placebo
- Cohort 1: GDC-0853 Placebo + Adalimumab Placebo (Placebo Comparator): Participants of Cohort 1 will receive placebo matched to GDC-0853, orally once daily along with placebo matched to adalimumab, subcutaneously Q2W starting on Day 1 for 12 weeks. Participants will remain on a stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week are allowed only if there is clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigator's discretion.
  Interventions: Drug: Folic Acid; Drug: MTX; Drug: Placebo
- Cohort 2: GDC-0853 High Dose (Experimental): Participants of Cohort 2 will receive GDC-0853 high dose, orally twice daily for 12 weeks. Participants will remain on a stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week are allowed only if there is clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigator's discretion.
  Interventions: Drug: GDC-0853; Drug: Folic Acid; Drug: MTX
- Cohort 2: GDC-0853 Placebo (Placebo Comparator): Participants of Cohort 2 will receive placebo matched to GDC-0853, orally twice daily for 12 weeks. Participants will remain on a stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week are allowed only if there is clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigator's discretion.
  Interventions: Drug: Folic Acid; Drug: MTX; Drug: Placebo

INTERVENTIONS:
Drug: GDC-0853 — Participants will receive GDC-0853 at low, mid, or high doses, orally once or twice daily for 12 weeks in Cohort 1 or 2.
  Other Names: RO7010939
  Arms: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo; Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo; Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo; Cohort 2: GDC-0853 High Dose
Drug: Adalimumab — Participants will receive adalimumab, subcutaneously Q2W starting on Day 1 for 12 weeks.
  Arms: Cohort 1: GDC-0853 Placebo + Adalimumab
Drug: Folic Acid — Participants will receive stable background therapy of folic acid of at least 5 mg total dose weekly (or equivalent) as per investigator's discretion.
Drug: MTX — Participants will receive stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week are allowed only if there is clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines).
Drug: Placebo — Participants will receive placebo matched to adalimumab, subcutaneously Q2W and/or placebo matched to GDC-0853, orally once or twice daily for 12 weeks in Cohort 1 or 2.
  Arms: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo; Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo; Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo; Cohort 1: GDC-0853 Placebo + Adalimumab; Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Cohort 2: GDC-0853 Placebo

SUMMARY:
This is a multicenter, Phase II, randomized, double-blind, placebo-controlled, active comparator (Cohort 1 only), parallel-group, dose-ranging study to evaluate the efficacy and safety of GDC-0853 in participants with moderate to severe active RA and an inadequate response to previous methotrexate (MTX) therapy (Cohort 1) or MTX and tumor necrosis factor (TNF) therapy who may have also had exposure to no more than one non-TNF inhibitor biologic (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of adult-onset RA as defined by the 2010 American College of Rheumatology/European League Against Rheumatism Classification Criteria for RA
* RA disease activity by joint counts and laboratory markers of inflammation: greater than or equal to (>=) 6 tender/painful joints on motion (68 joint count) and >= 6 swollen joints (66 joint count) at both screening and Day 1 (randomization)
* For MTX-inadequate response (IR) participants: must have had an inadequate response to MTX
* For TNF-IR participants: must have had an inadequate response or intolerance to previous treatment with at least 1 and no more than 2 biologic TNF-alpha inhibitors and may have also been exposed to no more than one biologic non-TNF-alpha inhibitor
* High sensitivity C-reactive protein of >= 0.400 milligrams per deciliter (mg/dL) for Cohort 1 and >= 0.650 mg/dL for Cohort 2 at screening

Exclusion Criteria:

* History of or current inflammatory joint disease other than RA or other systemic autoimmune disorder
* For MTX-IR participants: History of treatment with any TNF inhibitor, including biosimilar equivalents and history of treatment with biologic non-TNF-alpha inhibitor for RA
* For all participants: Previous treatment with cell-depleting therapy including B cell-depleting therapy (e.g., anti-cluster of differentiation 20-directed therapy such as rituximab), tofacitinib, or other Janus kinase inhibitor(s), or alkylating agents
* Current treatment with medications that are well known to prolong the QT interval at doses that have a clinically meaningful effect on QT
* History of non-gallstone-related pancreatitis or chronic pancreatitis
* Evidence of serious uncontrolled concomitant cardiac, neurologic, pulmonary, renal, hepatic, endocrine, metabolic, or gastrointestinal disease
* Evidence of chronic and/or active hepatitis B or C
* Women who are pregnant, nursing (breast feeding), or intending to become pregnant during the study or within 60 days after completion of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (150):
- United States (23):
  - Pinnacle Research Group; Llc, Central, Anniston, Alabama
  - Arizona Arthritis & Rheumatology Associates, P.C., Glendale, Arizona
  - Medvin Clinical Research, Covina, California
  - TriWest Research Associates, LLC, El Cajon, California
  - Saint Jude Heritage Medical Grp, Fullerton, California
  - Stanford University School of Medicine, Stanford, California
  - RASF-Clinical Research Center, Boca Raton, Florida
  - ZASA Clinical Research, Boynton Beach, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - InVentiv Health, Miami, Florida
  - Omega Research Consultants, Orlando, Florida
  - McIlwain Medical Group, Tampa, Florida
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - Medication Management, Greensboro, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Clinical Research Center of Reading, Wyomissing, Pennsylvania
  - Metroplex Clinical Research, Dallas, Texas
  - Baylor Research Inst., Dallas, Texas
  - Accurate Clinical Management - VO, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Crossroads Clinical Research, LLC, Victoria, Texas
  - Danville Orthopedic Clinic, Inc.; Research Department, Danville, Virginia
- Argentina (14):
  - Instituto de Investigaciones Clinicas-Mar del Plata, Buenos Aires
  - Organizacion Medica de Investigacion, Buenos Aires
  - Hospital Italiano, Buenos Aires
  - APRILLUS, Buenos Aires
  - Instituto centenario, Buenos Aires
  - Centro de Investigacion en Enfermedades Reumaticas CIER, Ciudad Autonoma Buenos Aires
  - Expertia S.A- Mautalen Salud e Investigación, Ciudad Autonoma Buenos Aires
  - CCBR - Buenos Aires - AR; AxisMed SRL, Ciudad Autonoma Buenos Aires
  - ILAIM-CEOM Inst. Latinoamericano de Inv. Medicas, Córdoba
  - Hospital Italiano de La Plata, La Plata
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Instituto de Investigaciones Clínicas Quilmes, Quilmes
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
  - Centro Medico Privado de Reumatologia; Reumathology, San Miguel
- Brazil (12):
  - CIP - Centro Internacional de Pesquisa; Pesquisa Clinica, Goiânia, Goiás
  - Centro Mineiro de Pesquisa - CMIP, Juiz de Fora, Minas Gerais
  - Edumed - Educação e Saúde SA, Curitiba, Paraná
  - Centro de Estudos em Terapias Inovadoras - CETI, Curtiba, Paraná
  - CCBR - Synarc Centro de Pesquisa Clinica - RJ, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - LMK Serviços Médicos S/S, Porto Alegre, Rio Grande do Sul
  - CAEP - Centro Avancado de Estudos e Pesquisas Ltda., Campinas, São Paulo
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas Ltda.; Pesquisa Clinica, São Paulo, São Paulo
  - Instituto de Pesquisa Clínica e Medicina Avançada Ltda, São Paulo, São Paulo
- Bulgaria (14):
  - MHAT - Dobrich, AD, Dobrich
  - MHAT "Eurohospital" - Plovdiv, OOD, Plovdiv
  - MHAT Kaspela; EOOD, Plovdiv
  - MHAT - Ruse, AD, Rousse
  - Medizinski Zentrar-1-Sevlievo EOOD, Sevlievo
  - MHAT "Hadzhi Dimitar", OOD, Sliven
  - Medical Center Excelsior OOD, Sofia
  - NMTH "Tsar Boris III", Sofia
  - MHAT "Lyulin", EAD, Sofia
  - DCC "Alexandrovska", EOOD; Clinic of Neurology, Sofia
  - UMHAT "SofiaMed", OOD, Sofia
  - MC "Synexus - Sofia", EOOD, Sofia
  - MHAT Dr. St. Kirkovich, AD, Stara Zagora
  - 'New Medical Center' , EOOD, Vratsa
- Colombia (6):
  - Centro de Reumatologia y Ortopedia, Barranquilla
  - Centro de Investigacion en Reumatologia y Especialdades Medicas SAS. CIREEM, Bogotá
  - Riesgo de Fractura S.A., Bogotá
  - Fundación Instituto de Reumatología Fernando Chalem, Bogotá
  - Clinica de Artritis Temprana S.A., Cali
  - Hospital Pablo Tobon Uribe, Medellín
- Mexico (9):
  - Consultorio Medico en Fundacion el Hospitalito de morelos A.C., Cuernavaca, Morelos
  - Centro de Investigación de Tratamientos Innovadores de Sinaloa (CITI), Culiacán, Sinaloa
  - Centro de Investigacion en Reumatologia, Mérida, Yucatán
  - Consultorio Particular del Dr. Miguel Cortes Hernandez, Cuernavaca
  - Centro de Investigacion en Enfermedades Reumaticas y Osteoporosis, Mexicali
  - Centro de Investigacion Clínica GRAMEL S.C, México
  - Policilinica Medica de Queretaro; Rheumatology, Querétaro
  - Clinical Research Institute, Tlalnepantla
  - Unidad de Enfermedades Reumaticas y Cronicodegenerativas, Torreón
- Poland (12):
  - NZOZ OSTEO-MEDIC S.C. Artur Racewicz, Jerzy Supronik, Bialystok
  - Szpital Uniwersytecki; nr 2 im. Dr J. Biziela, Bydgoszcz
  - Medica Pro Familia Spolka Akcyjna Oddzial w Katowicach, Katowice
  - Centrum Medyczne Plejady, Krakow
  - CCBR - Lodz - PL, Lodz
  - ETYKA Osrodek Badan Kliniczynch, Olsztyn
  - Ai Centrum Medyczne Sp. Z O.O Sp.K., Poznan
  - KO-MED Centra Kliniczne Staszow, Staszów
  - Medycyna Kliniczna, Warsaw
  - Centrum Medyczne AMED, Warsaw
  - Wojewódzki Szpital Specjalistyczny we Wrocławiu, Wroclaw
  - KO-MED Centra Kliniczne Zamosc, Zamość
- Russia (23):
  - TSBIH "Krasnoyarsk Interdistrict Clinical Hospital of Emergency Medical Care n.a. N.S. Karpovich, Krasnoyarsk, Krasnoyarsk Krai
  - Federal State Budgetary Scientific Institution Research Institute of Rheumatology V.A. Nasonova, Moscow, Moscow Oblast
  - SBIH of Moscow "City Clinical Hospital # 1 n. a. N. I. Pirogov", Moscow, Moscow Oblast
  - SBEI HPE " First Moscow State Medical University n.a. I.M. Sechenov" of the MoH of the RF, Moscow, Moscow Oblast
  - Technologii zdorovia LLC, Saint Petersburg, Sankt-Peterburg
  - Sanavita LLC, Saint Petersburg, Sankt-Peterburg
  - LLC Medical Sanitary Unit, Saint Petersburg, Sankt-Peterburg
  - Center of Family Medicine LC, Yekaterinburg, Sankt-Peterburg
  - SBHI of Yaroslavl Region Clinical Hospital #3, Yaroslavl, Volgograd Oblast
  - SMMIH "Chelyabinsk Regional Clinical Hospital", Chelyabinsk, Voronez
  - SAHI of Kem. "Regional Clinical Hospital for War Veterans", Kemerovo
  - OOO Family Polyclinic, Korolev, Moscow Region
  - Practical Medicine, Moscow
  - Limited Liability Company "Centre of Medical Common Practice", Novosibirsk
  - Ultramed, Omsk
  - City Hospital 25; Rheumatology, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - SBEI HPE "Saratov State Medical University n.a. V. I. Razumovskiy" of the MoH of the RF, Saratov
  - SBEI HPE "Smolensk State Medical University" of the MoH of the RF, Smolensk
  - Siberian State Medical University, Tomsk
  - SHI Ulyanovsk Reg Clinical Hospital, Ulyanovsk
  - Territorial Clinical Hospital #2, Vladivostok
  - SHI Yaroslavl Regional Clinical Hospital, Yaroslavl
- Serbia (6):
  - Institute of Rheumatology, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Institute of Treatment and Rehabilitation "Niska Banja", Niška Banja
  - Special hospital for rheumatic diseases Novi Sad, Novi Sad
  - General Hospital Sabac; Department of Urology and Hemodialysis, Šabac
- South Korea (7):
  - Chungnam National University Hospital; Department of Internal Medicine (Rheumatology), Daejeon
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center - Oncology, Seoul
  - Ajou University Hospital, Suwon
- Ukraine (24):
  - CI of TRC, Ternopil, Kherson Governorate
  - Regional CH Dep of Rheumatology SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk, KIEV Governorate
  - Medical Center Medical Clinic Blagomed LLC., Kyiv, KIEV Governorate
  - Medical Center OK!Clinic+, Kyiv, KIEV Governorate
  - SI NSС M.D. Strazhesko Institute of Cardiology of NAMSU, Kyiv, KIEV Governorate
  - Clinic of Modern Rheumatology Revmotsentr LLC, Kyiv, KIEV Governorate
  - Lviv Regional Clinical Hospital Dept of Rehmuaatology D. Halytskyi Lviv NMU, Lviv, KIEV Governorate
  - CH of State Border Service of Ukraine (Military Base 2522); Dept of Therapy, D.Halytskyi Lviv NMU, Lviv, KIEV Governorate
  - A.Novak Transcarpathian Regional Clinical Hospital, Uzhhorod, KIEV Governorate
  - Railway Transp DCH of HealthCenter Branch of PJSC Ukr Railway Dept of Rheumatology, Dnipro, Tavria Okruha
  - GI L.T.Malaya Therapy National Institute of the NAMS of Ukraine, Kharkiv
  - Kharkiv MA of PGE of MOHU Ch of Cardiology and Functional Diagnostics, Kharkiv
  - CNI Consultative and Diagnostic Center of Desnianskyi District of Kyiv, Kyiv
  - MI of Helathcare Kyiv RCH P.L. Shupy NMA of PGE, Kyiv
  - Gerontology Institute of the Ukrainian AMS, Kyiv
  - Oleksandrivska Clinical Hospital, Kyiv
  - Volyn Regional Center of Cardiovascular Pathology and Thrombolysis, Lutsk
  - City Hospital #1, Mykolaiv
  - M.V. Sklifosovsky Poltava RCH Dept of Rheumatology HSEIU UMSA, Poltava
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - M.I. Pyrogov VRCH Dept of Gastroenterology M.I. Pyrogov VNMU, Vinnytsia
  - City Clinical Hospital #9 Dept of Gastrosurgery SI Zaporizhzhia MA of PGE of MoHU, Zaporizhzhia
  - CI City Hospital #7, Zaporizhzhia
  - CI Zaporizhzhia Regional Clinical Hospital of ZRC, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 578 participants were enrolled in the study and 578 were dosed. One (1) subject in Cohort 2 in the Placebo arm was incorrectly dosed with the High Dose. The ITT data set included participants according to their randomization while SAF data set included participants according to the treatment administered.
Groups:
- Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo: Participants of Cohort 1 received GDC-0853 low dose, orally once daily along with placebo matched to adalimumab, subcutaneously Q2W starting on Day 1 for 12 weeks. Participants remained on a stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week are allowed only if there was clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigators discretion.
- Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo: Participants of Cohort 1 received GDC-0853 mid dose, orally twice daily along with placebo matched to adalimumab, subcutaneously Q2W starting on Day 1 for 12 weeks. Participants remained on a stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week were allowed only if there was clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigators discretion.
- Cohort 1: GDC-0853 High Dose + Adalimumab Placebo: Participants of Cohort 1 received GDC-0853 high dose, orally once daily along with placebo matched to adalimumab, subcutaneously every 2 weeks (Q2W) starting on Day 1 for 12 weeks. Participants remained on a stable background therapy of MTX 15-25 milligrams per week (mg/week) (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week were allowed only if there was clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigators discretion.
- Cohort 1: GDC-0853 Placebo + Adalimumab Placebo: Participants of Cohort 1 received placebo matched to GDC-0853, orally once daily along with placebo matched to adalimumab, subcutaneously Q2W starting on Day 1 for 12 weeks. Participants remained on a stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week were allowed only if there was clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigators discretion.
- Cohort 1: GDC-0853 Placebo + Adalimumab: Participants of Cohort 1 received placebo matched to GDC-0853, orally once daily along with adalimumab, subcutaneously Q2W starting on Day 1 for 12 weeks. Participants remained on a stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week were allowed only if there was clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigators discretion.
- Cohort 2: GDC-0853 High Dose: Participants of Cohort 2 received GDC-0853 high dose, orally twice daily for 12 weeks. Participants remained on a stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week were allowed only if there was clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigators discretion.
- Cohort 2: GDC-0853 Placebo: Participants of Cohort 2 received placebo matched to GDC-0853, orally twice daily for 12 weeks. Participants remained on a stable background therapy of MTX 15-25 mg/week (oral or parenteral; for participants entering the trial on MTX doses 15 mg/week, doses as low as 7.5 mg/week were allowed only if there was clear documentation in the medical record that higher doses were not tolerated or that the dose of MTX is the highest acceptable dose based on local clinical practice guidelines) and folic acid of at least 5 mg total dose weekly (or equivalent) as per investigators discretion.
Period: Overall Study
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Started (SAF population) | 40 | 109 | 110 | 110 | 111 | 49 | 49
Randomized (ITT population) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Completed | 37 | 100 | 102 | 102 | 108 | 48 | 44
Not Completed | 3 | 9 | 8 | 8 | 3 | 1 | 5
Not completed — Adverse Event | 0 | 3 | 4 | 4 | 1 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 2 | 1 | 4 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3 | 2 | 0 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population (SAF) included all subjects that received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo | Total
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 49 | 49 | 578
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 95 | 99 | 98 | 98 | 41 | 40 | 506
  >=65 years | 5 | 14 | 11 | 12 | 13 | 8 | 9 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.3 (12.0) | 50.4 (11.0) | 49.9 (12.4) | 50.2 (11.6) | 49.9 (12.4) | 51.3 (13.2) | 54.6 (11.5) | 50.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 92 | 85 | 90 | 87 | 37 | 37 | 463
  Male | 5 | 17 | 25 | 20 | 24 | 12 | 12 | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    American Indian or Alaska native | 0 | 8 | 12 | 11 | 9 | 6 | 5 | 51
    Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Black of African American | 0 | 1 | 2 | 3 | 1 | 1 | 2 | 10
    White | 36 | 96 | 96 | 95 | 99 | 42 | 42 | 506
    Multiple | 3 | 2 | 0 | 1 | 1 | 0 | 0 | 7
    Unknown | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 8 | 38 | 40 | 38 | 39 | 17 | 15 | 195
    Not Hispanic or Latino | 31 | 68 | 69 | 72 | 70 | 32 | 33 | 375
    Not Stated | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3
    Unknown | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Day 84, Comparison Between GDC-0853 and Placebo (Cohort 1)
Description: ACR50 response is defined as a ≥ 50% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Day 84
Population: Intent-to-Treat (ITT) All randomized participants who received any part of an infusion of study medication were included in the ITT analysis. Number of participants for whom data were collected is indicated for each time point.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111
Percentage | 17.5 [5.72 to 29.28] | 27.5 [19.14 to 35.91] | 34.5 [25.66 to 43.43] | 14.5 [7.96 to 21.13] | 36.0 [27.10 to 44.97]
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Test type: Superiority; p = 0.2503, Cochran-Mantel-Haenszel; Weighted difference = 8.00, 95% CI 2-sided [-5.64 to 21.64]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Test type: Superiority; p = 0.0164, Cochran-Mantel-Haenszel; Weighted difference = 12.93, 95% CI 2-sided [2.37 to 23.48]
Statistical Analysis 3: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Weighted difference = 20.00, 95% CI 2-sided [9.21 to 30.79]

2. Primary Outcome: Percentage of Participants With Adverse Events
Description: An Adverse event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events. A SAE was any experience that suggested a significant hazard, contraindication, side effect or precaution that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant.
Time Frame: Day 1 up to 8 weeks after last dose (up to Week 20)
Population: Safety population included all participants according to treatment administered.
Measure: Number; unit: Percentage
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 49 | 49
Percentage | 37.5 | 42.2 | 50.9 | 45.5 | 45.0 | 22.4 | 44.9

3. Secondary Outcome: Percentage of Participants Achieving ACR50 Response at Day 84, Comparison Between GDC-0853 and Adalimumab (Cohort 1)
Description: as for outcome 1
Time Frame: Day 84
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111
Percentage | 17.5 [5.72 to 29.28] | 27.5 [19.14 to 35.91] | 34.5 [25.66 to 43.43] | 14.5 [7.96 to 21.13] | 36.0 [27.10 to 44.97]
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Test type: Superiority; p = 0.1694, Cochran-Mantel-Haenszel; Weighted difference = -8.58, 95% CI 2-sided [-20.82 to 3.66]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Test type: Superiority; p = 0.8132, Cochran-Mantel-Haenszel; Weighted difference = -1.50, 95% CI [-13.96 to 10.95]

4. Secondary Outcome: Percentage of Participants Achieving ACR50 Response at Day 84, Comparison Between GDC-0853 and Placebo (Cohort 2)
Description: as for outcome 1
Time Frame: Day 84
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 48 | 50
Percentage | 25.0 [12.75 to 37.25] | 12.0 [2.99 to 21.01]
Statistical Analysis 1: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Test type: Superiority; p = 0.0717, Cochran-Mantel-Haenszel; Weighted difference = 13.7, 95% CI 2-sided [-1.21 to 28.61]

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response is defined as a ≥ 20% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate]
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Percentage
  Week 1 Day 7 | 10.0 [.70 to 19.3] | 14.7 [8.04 to 21.32] | 13.6 [7.22 to 20.05] | 10.0 [4.39 to 15.61] | 25.2 [17.15 to 33.30] | 22.9 [11.03 to 34.81] | 2.0 [0.00 to 5.88]
  Week 2 Day 14 | 12.5 [2.25 to 22.75] | 19.3 [11.86 to 26.67] | 27.3 [18.95 to 35.60] | 16.4 [9.45 to 23.28] | 48.6 [39.35 to 57.95] | 25.0 [12.75 to 37.25] | 10.0 [1.68 to 18.32]
  Week 4 Day 28 | 30.0 [15.80 to 44.20] | 34.9 [25.92 to 43.81] | 41.8 [32.60 to 51.04] | 25.5 [17.31 to 33.59] | 59.5 [50.33 to 68.59] | 35.4 [21.89 to 48.95] | 24.0 [12.16 to 35.84]
  Week 8 Day 56 | 50.0 [34.51 to 65.49] | 52.3 [42.92 to 61.67] | 58.2 [48.96 to 67.40] | 37.3 [28.24 to 46.31] | 71.2 [62.74 to 79.60] | 47.9 [33.78 to 62.05] | 18.0 [7.35 to 28.65]
  Week 12 Day 84 | 60.0 [44.82 to 75.18] | 56.0 [46.64 to 65.28] | 59.1 [49.90 to 68.28] | 36.4 [27.37 to 45.35] | 72.1 [63.73 to 80.42] | 58.3 [44.39 to 72.28] | 24.0 [12.16 to 35.84]

6. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: as for outcome 1
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Percentage
  Week 1 Day 7 | 2.5 [0.00 to 7.34] | 2.8 [0.00 to 5.82] | 3.6 [0.14 to 7.13] | 2.7 [0.00 to 5.77] | 4.5 [0.65 to 8.36] | 6.3 [0.00 to 13.10] | 2.0 [0.00 to 5.88]
  Week 2 Day 14 | 0.0 [0.00 to 0.00] | 1.8 [0.00 to 4.35] | 7.3 [2.42 to 12.13] | 2.7 [0.00 to 5.77] | 9.0 [3.68 to 14.34] | 10.4 [1.77 to 19.06] | 0.00 [0.00 to 0.00]
  Week 4 day 28 | 5.0 [0.00 to 11.75] | 9.2 [3.76 to 14.59] | 10.0 [4.39 to 15.61] | 6.4 [1.80 to 10.93] | 25.2 [17.15 to 33.30] | 10.4 [1.77 to 19.06] | 6.0 [0.00 to 12.58]
  Week 8 Day 56 | 15.0 [3.93 to 26.07] | 18.3 [11.08 to 25.62] | 22.7 [14.9 to 30.56] | 17.3 [10.21 to 24.34] | 32.4 [23.72 to 41.14] | 22.9 [11.03 to 34.81] | 10.0 [1.68 to 18.32]
  Week 12 Day 84 | 17.5 [5.72 to 29.28] | 27.5 [19.14 to 35.91] | 34.5 [25.66 to 43.43] | 14.5 [7.96 to 21.13] | 36.0 [27.10 to 44.97] | 25.0 [12.75 to 37.25] | 12.0 [2.99 to 21.01]

7. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response is defined as a ≥ 70% improvement (reduction) compared with Baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Percentage
  Week 1 Day 7 | 0.0 [0.00 to 0.00] | 0.9 [0.00 to 2.71] | 0.9 [0.00 to 2.68] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Week 2 Day 14 | 0.0 [0.00 to 0.00] | 0.9 [0.00 to 2.71] | 0.0 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 3.6 [0.14 to 7.07] | 4.2 [0.00 to 9.82] | 0.0 [0.00 to 0.00]
  Week 4 Day 28 | 0 [0.00 to 0.00] | 2.8 [0.00 to 5.82] | 4.5 [0.65 to 8.44] | 0.9 [0.00 to 2.68] | 6.3 [1.78 to 10.83] | 2.1 [0.00 to 6.12] | 2.0 [0.00 to 5.88]
  Week 8 Day 56 | 0.0 [0.00 to 0.00] | 7.3 [2.44 to 12.24] | 9.1 [3.72 to 14.46] | 3.6 [0.14 to 7.13] | 14.4 [7.88 to 20.95] | 6.3 [0.00 to 13.10] | 4.0 [0.00 to 9.43]
  Week 12 Day 84 | 5.0 [0.00 to 11.75] | 9.2 [3.76 to 14.59] | 12.7 [6.50 to 18.96] | 7.3 [2.42 to 12.13] | 18.0 [10.87 to 25.17] | 14.6 [4.60 to 24.57] | 4.0 [0.00 to 9.43]

8. Secondary Outcome: Change in Disease Activity Score From Baseline Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP])
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. DAS28 Remission is defined as a DAS28 score < 2.6.
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale
  Week 1 Day 7: number analyzed (Participants) | 37 | 106 | 107 | 109 | 107 | 47 | 46
  Week 1 Day 7 | -0.34 (0.60) | -0.35 (0.66) | -0.37 (0.80) | -0.33 (0.84) | -0.92 (0.71) | -0.49 (0.84) | -0.36 (0.63)
  Week 2 Day 14: number analyzed (Participants) | 38 | 106 | 108 | 110 | 109 | 48 | 47
  Week 2 Day 14 | -0.47 (0.72) | -0.63 (0.84) | -0.70 (0.80) | -.54 (0.90) | -1.09 (0.81) | -0.65 (0.87) | -0.45 (0.69)
  Week 4 Day 28: number analyzed (Participants) | 37 | 103 | 105 | 105 | 109 | 47 | 48
  Week 4 Day 28 | -0.75 (0.86) | -0.90 (0.96) | -0.91 (0.97) | -0.62 (1.04) | -1.45 (0.87) | -0.77 (0.90) | -0.44 (0.84)
  Week 8 Day 56: number analyzed (Participants) | 36 | 100 | 103 | 100 | 106 | 47 | 45
  Week 8 Day 56 | -1.14 (0.90) | -1.35 (1.12) | -1.37 (1.11) | -1.08 (1.19) | -1.75 (0.98) | -1.33 (0.98) | -0.56 (0.87)
  Week 12 Day 84: number analyzed (Participants) | 37 | 97 | 97 | 102 | 106 | 47 | 44
  Week 12 Day 84 | -1.30 (0.95) | -1.72 (1.11) | -1.70 (1.02) | -1.17 (1.24) | -1.87 (1.02) | -1.62 (1.15) | -0.86 (1.03)
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.8504, ANCOVA; adjusted difference = -0.11, 95% CI 2-sided [-0.45 to 0.23]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; At week 1, Day 7; Test type: Superiority; p = 0.9884, ANCOVA; Adjusted Difference = -0.04, 95% CI 2-sided [-0.28 to 0.21]
Statistical Analysis 3: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1 Day 7; Test type: Superiority; p = 0.9230, ANCOVA; Adjusted Difference = -0.06, 95% CI 2-sided [-0.31 to 0.18]
Statistical Analysis 4: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.9853, ANCOVA; Adjusted Difference = -0.06, 95% CI 2-sided [-0.43 to 0.31]
Statistical Analysis 5: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.6826, ANCOVA; Adjusted Difference = -0.12, 95% CI 2-sided [-0.38 to 0.15]
Statistical Analysis 6: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.2634, ANCOVA; Adjusted Difference = -0.18, 95% CI 2-sided [-0.45 to 0.08]
Statistical Analysis 7: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.2885, ANCOVA; Adjusted Difference = -0.29, 95% CI 2-sided [-0.72 to 0.14]
Statistical Analysis 8: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0598, ANCOVA; Adjusted Difference = -0.30, 95% CI 2-sided [-0.61 to 0.01]
Statistical Analysis 9: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0440, ANCOVA; Adjusted Difference = -0.31, 95% CI 2-sided [-0.62 to -0.01]
Statistical Analysis 10: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.4271, ANCOVA; Adjusted Difference = -0.28, 95% CI 2-sided [-0.76 to 0.20]
Statistical Analysis 11: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.0969, ANCOVA; Adjusted Difference = -0.31, 95% CI 2-sided [-0.66 to 0.04]
Statistical Analysis 12: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.0612, ANCOVA; Adjusted Difference = -0.33, 95% CI 2-sided [-0.68 to 0.01]
Statistical Analysis 13: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.2079, ANCOVA; Adjusted Difference = -0.36, 95% CI 2-sided [-0.84 to 0.12]
Statistical Analysis 14: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0003, ANCOVA; Adjusted Difference = -0.57, 95% CI 2-sided [-0.92 to -0.22]
Statistical Analysis 15: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0003, ANCOVA; Adjusted Difference = -0.57, 95% CI 2-sided [-0.92 to -0.22]
Statistical Analysis 16: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 1, Day 7; Test type: Superiority; p < .0001, ANCOVA; Adjusted Difference = 0.58, 95% CI 2-sided [0.34 to 0.82]
Statistical Analysis 17: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 1, Day 7; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Net) = 0.55, 95% CI 2-sided [0.31 to 0.80]
Statistical Analysis 18: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 2, Day 14; Test type: Superiority; p < .0001, ANCOVA; Adjusted Difference = 0.47, 95% CI 2-sided [0.20 to 0.74]
Statistical Analysis 19: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 2, Day 14; Test type: Superiority; p = 0.0009, ANCOVA; Adjusted Difference = 0.40, 95% CI 2-sided [0.13 to 0.66]
Statistical Analysis 20: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 4, Day 28; Test type: Superiority; p < .0001, ANCOVA; Adjusted Difference = 0.56, 95% CI 2-sided [0.25 to 0.87]
Statistical Analysis 21: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 4, Day 28; Test type: Superiority; p < .0001, ANCOVA; Adjusted Difference = 0.55, 95% CI 2-sided [0.24 to 0.85]
Statistical Analysis 22: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 8, Day 56; Test type: Superiority; p = 0.0095, ANCOVA; Adjusted Difference = 0.42, 95% CI 2-sided [0.08 to 0.76]
Statistical Analysis 23: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 8, Day 56; Test type: Superiority; p = 0.0153, ANCOVA; Adjusted Difference = 0.40, 95% CI 2-sided [0.06 to 0.74]
Statistical Analysis 24: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 12, Day 84; Test type: Superiority; p = 0.4839, ANCOVA; Adjusted Difference = 0.19, 95% CI 2-sided [-0.16 to 0.54]
Statistical Analysis 25: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 12, Day 84; Test type: Superiority; p = 0.5035, ANCOVA; Adjusted Difference = 0.19, 95% CI 2-sided [-0.16 to 0.53]
Statistical Analysis 26: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 1, Day 7; Test type: Superiority; p = 0.4286, ANCOVA; Adjusted Difference = -0.11, 95% CI 2-sided [-0.38 to 0.16]
Statistical Analysis 27: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 2, Day 14; Test type: Superiority; p = 0.1831, ANCOVA; Adjusted Difference = -0.20, 95% CI 2-sided [-0.50 to 0.10]
Statistical Analysis 28: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0667, ANCOVA; Adjusted Difference = -0.31, 95% CI 2-sided [-0.65 to 0.02]
Statistical Analysis 29: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 8, Day 56; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted Difference = -0.77, 95% CI 2-sided [-1.11 to -0.42]
Statistical Analysis 30: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0002, ANCOVA; Adjusted Difference = -0.76, 95% CI 2-sided [-1.15 to -0.38]

9. Secondary Outcome: Change in Disease Activity Score From Baseline Based on 28-Joints Count and C-Reactive Protein (4 Variables) (DAS28-4 [CRP])
Description: as for outcome 8
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale
  Week 1 Day 7: number analyzed (Participants) | 37 | 104 | 102 | 103 | 104 | 47 | 45
  Week 1 Day 7 | -0.43 (0.67) | -0.48 (0.73) | -0.49 (0.86) | -0.37 (0.91) | -1.10 (0.75) | -0.63 (0.91) | -.40 (0.69)
  Week 2 Day 14: number analyzed (Participants) | 37 | 103 | 105 | 105 | 107 | 48 | 46
  Week 2 Day 14 | -0.51 (0.85) | -0.77 (0.86) | -0.84 (0.86) | -0.57 (1.00) | -1.26 (0.89) | -0.81 (0.98) | -0.54 (0.80)
  Week 4 Day 28: number analyzed (Participants) | 36 | 101 | 103 | 99 | 106 | 47 | 48
  Week 4 Day 28 | -0.88 (0.90) | -1.06 (1.02) | -1.08 (1.03) | -0.65 (1.16) | -1.61 (0.94) | -0.95 (1.04) | -0.55 (0.94)
  Week 8 Day 56: number analyzed (Participants) | 36 | 99 | 100 | 97 | 103 | 47 | 45
  Week 8 Day 56 | -1.31 (0.91) | -1.56 (1.21) | -1.57 (1.16) | 1.20 (1.30) | -1.97 (1.03) | -1.51 (1.05) | -0.67 (1.01)
  Week 12 Day 84: number analyzed (Participants) | 36 | 94 | 95 | 99 | 104 | 47 | 43
  Week 12 Day 84 | -1.53 (0.95) | -1.97 (1.20) | -1.93 (1.11) | -1.33 (1.33) | -2.06 (1.08) | -1.83 (1.22) | -1.00 (1.11)
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.5807, ANCOVA; Adjusted Difference = -0.18, 95% CI 2-sided [-0.55 to 0.19]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.6270, ANCOVA; Adjusted Difference = -0.12, 95% CI 2-sided [-0.39 to 0.14]
Statistical Analysis 3: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.4475, ANCOVA; Adjusted Difference = -0.15, 95% CI 2-sided [-0.42 to 0.12]
Statistical Analysis 4: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.9891, ANCOVA; Adjusted Difference = -0.06, 95% CI 2-sided [-0.47 to 0.35]
Statistical Analysis 5: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.2244, ANCOVA; Adjusted Difference = -0.21, 95% CI 2-sided [-0.51 to 0.08]
Statistical Analysis 6: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.0586, ANCOVA; Adjusted Difference = -0.28, 95% CI 2-sided [-0.58 to 0.01]
Statistical Analysis 7: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.1338, ANCOVA; Adjusted Difference = -0.39, 95% CI 2-sided [-0.85 to 0.08]
Statistical Analysis 8: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0119, ANCOVA; Adjusted Difference = -0.40, 95% CI 2-sided [-0.74 to -0.07]
Statistical Analysis 9: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0046, ANCOVA; Adjusted Difference = -0.44, 95% CI 2-sided [-0.77 to -0.11]
Statistical Analysis 10: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.3943, ANCOVA; Adjusted Difference = -0.31, 95% CI 2-sided [-0.82 to 0.20]
Statistical Analysis 11: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.0526, ANCOVA; Adjusted Difference = -0.37, 95% CI 2-sided [-0.74 to 0.00]
Statistical Analysis 12: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.0365, ANCOVA; Adjusted Difference = -0.39, 95% CI 2-sided [-0.76 to -0.02]
Statistical Analysis 13: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.1696, ANCOVA; Adjusted Difference = -0.41, 95% CI 2-sided [-0.93 to 0.11]
Statistical Analysis 14: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0002, ANCOVA; Adjusted Difference = -0.63, 95% CI 2-sided [-1.01 to -0.25]
Statistical Analysis 15: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0003, ANCOVA; Adjusted Difference = -0.62, 95% CI 2-sided [-1.00 to -0.24]
Statistical Analysis 16: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 1, Day 7; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted Difference = 0.64, 95% CI 2-sided [0.37 to 0.90]
Statistical Analysis 17: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 1, Day 7; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted Difference = 0.61, 95% CI 2-sided [0.34 to 0.88]
Statistical Analysis 18: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 2, Day 14; Test type: Superiority; p = 0.0001, ANCOVA; Adjusted Difference = 0.50, 95% CI 2-sided [0.21 to 0.79]
Statistical Analysis 19: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 2, Day 14; Test type: Superiority; p = 0.0012, ANCOVA; Adjusted Difference = 0.43, 95% CI 2-sided [0.14 to 0.72]
Statistical Analysis 20: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 4, Day 28; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted Difference = 0.58, 95% CI 2-sided [0.25 to 0.91]
Statistical Analysis 21: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 4, Day 28; Test type: Superiority; p = 0.0002, ANCOVA; Adjusted Difference = 0.54, 95% CI 2-sided [0.21 to 0.87]
Statistical Analysis 22: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 8, Day 56; Test type: Superiority; p = 0.0084, ANCOVA; Adjusted Difference = 0.46, 95% CI 2-sided [0.09 to 0.82]
Statistical Analysis 23: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 8, Day 56; Test type: Superiority; p = 0.0124, ANCOVA; Adjusted Difference = 0.44, 95% CI 2-sided [0.07 to 0.80]
Statistical Analysis 24: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 12, Day 84; Test type: Superiority; p = 0.7565, ANCOVA; Adjusted Difference = 0.15, 95% CI 2-sided [-0.23 to 0.52]
Statistical Analysis 25: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 12, Day 84; Test type: Superiority; p = 0.7158, ANCOVA; Adjusted Difference = 0.16, 95% CI 2-sided [-0.22 to 0.53]
Statistical Analysis 26: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 1, Day 7; Test type: Superiority; p = 0.1368, ANCOVA; Adjusted Difference = -0.22, 95% CI 2-sided [-0.52 to 0.07]
Statistical Analysis 27: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 2, Day 14; Test type: Superiority; p = 0.0974, ANCOVA; Adjusted Difference = -0.28, 95% CI 2-sided [-0.62 to 0.05]
Statistical Analysis 28: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0479, ANCOVA; Adjusted Difference = -0.38, 95% CI 2-sided [-0.76 to -0.00]
Statistical Analysis 29: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 8, Day 56; Test type: Superiority; p < 0.0001, ANCOVA; Adjusted Difference = -0.84, 95% CI 2-sided [-1.22 to -0.46]
Statistical Analysis 30: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0001, ANCOVA; Adjusted Difference = -0.83, 95% CI 2-sided [-1.24 to -0.42]

10. Secondary Outcome: Change in Disease Activity Score From Baseline Based on 28-Joints Count and Erythrocyte Sedimentation Rate (3 Variables) (DAS28-3 [ESR])
Description: as for outcome 8
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale
  Week 1 Day 7: number analyzed (Participants) | 38 | 105 | 108 | 110 | 106 | 47 | 47
  Week 1 Day 7 | -0.35 (0.57) | -0.42 (0.65) | -0.39 (0.68) | -0.34 (0.86) | -0.72 (0.72) | -0.50 (0.73) | -0.31 (0.60)
  Week 2 Day 14: number analyzed (Participants) | 39 | 105 | 109 | 110 | 109 | 47 | 48
  Week 2 Day 14 | -0.60 (0.89) | -0.69 (0.84) | -0.68 (0.74) | -0.55 (0.92) | -1.02 (0.84) | -0.64 (0.81) | -0.51 (0.73)
  Week 4 Day 28: number analyzed (Participants) | 38 | 104 | 106 | 108 | 109 | 47 | 48
  Week 4 Day 28 | -0.88 (0.89) | -0.99 (0.98) | -0.97 (0.90) | -0.75 (1.02) | -1.47 (1.02) | -0.85 (0.81) | -0.50 (0.83)
  Week 8 Day 56: number analyzed (Participants) | 37 | 100 | 103 | 102 | 108 | 47 | 45
  Week 8 Day 56 | -1.25 (0.85) | -1.44 (1.14) | -1.40 (1.06) | -1.15 (1.19) | -1.74 (0.98) | -1.35 (0.96) | -0.70 (0.98)
  Week 12 Day 84: number analyzed (Participants) | 37 | 97 | 97 | 102 | 108 | 47 | 45
  Week 12 Day 84 | -1.51 (1.01) | -1.80 (1.25) | -1.80 (0.99) | -1.30 (1.22) | -1.85 (1.06) | -1.65 (1.06) | -0.94 (10.6)
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.9193, ANCOVA; Adjusted Difference = -0.09, 95% CI 2-sided [-0.41 to 0.24]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.7062, ANCOVA; Adjusted Difference = -0.10, 95% CI 2-sided [-0.33 to 0.14]
Statistical Analysis 3: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.8542, ANCOVA; Adjusted Difference = -0.08, 95% CI 2-sided [-0.31 to 0.16]
Statistical Analysis 4: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.8095, ANCOVA; Adjusted Difference = -0.13, 95% CI 2-sided [-0.51 to 0.24]
Statistical Analysis 5: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.3862, ANCOVA; Adjusted Difference = -0.17, 95% CI 2-sided [-0.44 to 0.11]
Statistical Analysis 6: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.4328, ANCOVA; Adjusted Difference = -0.16, 95% CI 2-sided [-0.43 to 0.12]
Statistical Analysis 7: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.4915, ANCOVA; Adjusted Difference = -0.24, 95% CI 2-sided [-0.68 to 0.20]
Statistical Analysis 8: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.1441, ANCOVA; Adjusted Difference = -0.26, 95% CI 2-sided [-0.58 to 0.06]
Statistical Analysis 9: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.1890, ANCOVA; Adjusted Difference = -0.24, 95% CI 2-sided [-0.56 to 0.07]
Statistical Analysis 10: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.5566, ANCOVA; Adjusted Difference = -0.25, 95% CI 2-sided [-0.74 to -0.24]
Statistical Analysis 11: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.0920, ANCOVA; Adjusted Difference = -0.32, 95% CI 2-sided [-0.68 to 0.04]
Statistical Analysis 12: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.1391, ANCOVA; Adjusted Difference = -0.29, 95% CI 2-sided [-0.65 to 0.06]
Statistical Analysis 13: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.2873, ANCOVA; Adjusted Difference = -0.35, 95% CI 2-sided [-0.86 to 0.17]
Statistical Analysis 14: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0020, ANCOVA; Adjusted Difference = -0.54, 95% CI 2-sided [-0.91 to -0.16]
Statistical Analysis 15: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0016, ANCOVA; Adjusted Difference = -0.54, 95% CI 2-sided [-0.92 to -0.17]
Statistical Analysis 16: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 1, Day 7; Test type: Superiority; p = 0.0050, ANCOVA; Adjusted Difference = 0.31, 95% CI 2-sided [0.07 to 0.55]
Statistical Analysis 17: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 1, Day 7; Test type: Superiority; p = 0.0020, ANCOVA; Adjusted Difference = 0.33, 95% CI 2-sided [0.10 to 0.57]
Statistical Analysis 18: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 2, Day 14; Test type: Superiority; p = 0.0082, ANCOVA; Adjusted Difference = 0.35, 95% CI 2-sided [0.07 to 0.62]
Statistical Analysis 19: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 2, Day 14; Test type: Superiority; p = 0.0056, ANCOVA; Adjusted Difference = 0.35, 95% CI 2-sided [0.08 to 0.63]
Statistical Analysis 20: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 4, Day 28; Test type: Superiority; p = 0.0004, ANCOVA; Adjusted Difference = 0.50, 95% CI 2-sided [0.19 to 0.82]
Statistical Analysis 21: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 4, Day 28; Test type: Superiority; p = 0.0002, ANCOVA; Adjusted Difference = 0.52, 95% CI 2-sided [0.21 to 0.84]
Statistical Analysis 22: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 8, Day 56; Test type: Superiority; p = 0.0650, ANCOVA; Adjusted Difference = 0.34, 95% CI 2-sided [-0.01 to 0.69]
Statistical Analysis 23: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 8, Day 56; Test type: Superiority; p = 0.0365, ANCOVA; Adjusted Difference = 0.37, 95% CI 2-sided [0.02 to 0.72]
Statistical Analysis 24: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 12, Day 84; Test type: Superiority; p = 0.9338, ANCOVA; Adjusted Difference = 0.09, 95% CI 2-sided [-0.28 to 0.47]
Statistical Analysis 25: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 12, Day 84; Test type: Superiority; p = 0.9520, ANCOVA; Adjusted Difference = 0.09, 95% CI 2-sided [-0.29 to 0.46]
Statistical Analysis 26: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 1, Day 7; Test type: Superiority; p = 0.1496, ANCOVA; Adjusted Difference = -0.19, 95% CI 2-sided [-0.45 to 0.07]
Statistical Analysis 27: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 2, Day 14; Test type: Superiority; p = 0.3936, ANCOVA; Adjusted Difference = -0.13, 95% CI 2-sided [-0.43 to 0.17]
Statistical Analysis 28: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0346, ANCOVA; Adjusted Difference = -0.35, 95% CI 2-sided [-0.68 to -0.03]
Statistical Analysis 29: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 8, Day 56; Test type: Superiority; p = 0.0004, ANCOVA; Adjusted Difference = -0.68, 95% CI 2-sided [-1.04 to -0.31]
Statistical Analysis 30: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0003, ANCOVA; Adjusted Difference = -0.73, 95% CI 2-sided [-1.11 to -0.34]

11. Secondary Outcome: Change in Disease Activity Score From Baseline Based on 28-Joints Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 [ESR])
Description: as for outcome 8
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale
  Week 1 Day 7: number analyzed (Participants) | 38 | 103 | 103 | 104 | 103 | 47 | 45
  Week 1 Day 7 | -0.45 (0.63) | -0.54 (0.72) | -0.52 (0.77) | -0.37 (0.95) | -0.93 (0.76) | -0.65 (0.80) | -0.36 (0.66)
  Week 2 Day 14: number analyzed (Participants) | 38 | 102 | 106 | 105 | 107 | 47 | 47
  Week 2 Day 14 | -0.63 (0.98) | -0.85 (0.85) | -0.84 (0.82) | -0.58 (1.03) | -1.22 (0.94) | -0.81 (0.92) | -0.60 (0.84)
  Week 4 Day 28: number analyzed (Participants) | 37 | 102 | 104 | 102 | 106 | 47 | 48
  Week 4 Day 28 | -1.00 (0.95) | -1.16 (1.06) | -1.15 (0.98) | -0.79 (1.16) | -1.65 (1.11) | -1.04 (0.95) | -0.61 (0.96)
  Week 8 Day 56: number analyzed (Participants) | 37 | 99 | 100 | 99 | 105 | 47 | 45
  Week 8 Day 56 | -1.43 (0.88) | -1.67 (1.25) | -1.63 (1.14) | -1.29 (1.31) | -2.00 (1.06) | -1.54 (1.04) | -0.81 (1.12)
  Week 12 Day 84: number analyzed (Participants) | 36 | 94 | 95 | 99 | 106 | 47 | 44
  Week 12 Day 84 | -1.76 (1.04) | -2.06 (1.36) | -2.05 (1.08) | -1.46 (1.32) | -2.08 (1.14) | -1.89 (1.15) | -1.08 (1.17)
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.6083, ANCOVA; Adjusted Difference = -0.17, 95% CI 2-sided [-0.53 to 0.19]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.2672, ANCOVA; Adjusted Difference = -0.18, 95% CI 2-sided [-0.44 to 0.08]
Statistical Analysis 3: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.3158, ANCOVA; Adjusted Difference = -0.17, 95% CI 2-sided [-0.43 to 0.09]
Statistical Analysis 4: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.8495, ANCOVA; Adjusted Difference = -0.14, 95% CI 2-sided [-0.55 to 0.28]
Statistical Analysis 5: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.0856, ANCOVA; Adjusted Difference = -0.28, 95% CI 2-sided [-0.58 to 0.03]
Statistical Analysis 6: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.1021, ANCOVA; Adjusted Difference = -0.27, 95% CI 2-sided [-0.57 to 0.04]
Statistical Analysis 7: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.2762, ANCOVA; Adjusted Difference = -0.33, 95% CI 2-sided [-0.82 to 0.15]
Statistical Analysis 8: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0286, ANCOVA; Adjusted Difference = -0.38, 95% CI 2-sided [-0.73 to -0.03]
Statistical Analysis 9: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0274, ANCOVA; Adjusted Difference = -0.38, 95% CI 2-sided [-0.73 to -0.03]
Statistical Analysis 10: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.4981, ANCOVA; Adjusted Difference = -0.28, 95% CI 2-sided [-0.81 to 0.24]
Statistical Analysis 11: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.0472, ANCOVA; Adjusted Difference = -0.39, 95% CI 2-sided [-0.78 to -0.00]
Statistical Analysis 12: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.0753, ANCOVA; Adjusted Difference = -0.36, 95% CI 2-sided [-0.75 to 0.03]
Statistical Analysis 13: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.1853, ANCOVA; Adjusted Difference = -0.43, 95% CI 2-sided [-0.99 to 0.13]
Statistical Analysis 14: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0009, ANCOVA; Adjusted Difference = -0.62, 95% CI 2-sided [-1.03 to -0.21]
Statistical Analysis 15: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0008, ANCOVA; Adjusted Difference = -0.62, 95% CI 2-sided [-1.03 to -0.21]
Statistical Analysis 16: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 1, Day 7; Test type: Superiority; p = 0.0005, ANCOVA; Adjusted Difference = 0.41, 95% CI 2-sided [0.15 to 0.67]
Statistical Analysis 17: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 1, Day 7; Test type: Superiority; p = 0.0003, ANCOVA; Adjusted Difference = 0.42, 95% CI 2-sided [0.16 to 0.68]
Statistical Analysis 18: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 2, Day 14; Test type: Superiority; p = 0.0060, ANCOVA; Adjusted Difference = 0.39, 95% CI 2-sided [0.09 to 0.69]
Statistical Analysis 19: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 2, Day 14; Test type: Superiority; p = 0.0039, ANCOVA; Adjusted Difference = 0.40, 95% CI 2-sided [0.10 to 0.70]
Statistical Analysis 20: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 4, Day 28; Test type: Superiority; p = 0.0007, ANCOVA; Adjusted Difference = 0.53, 95% CI 2-sided [0.18 to 0.88]
Statistical Analysis 21: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 4, Day 28; Test type: Superiority; p = 0.0007, ANCOVA; Adjusted Difference = 0.53, 95% CI 2-sided [0.19 to 0.88]
Statistical Analysis 22: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 8, Day 56; Test type: Superiority; p = 0.0450, ANCOVA; Adjusted Difference = 0.39, 95% CI 2-sided [0.01 to 0.77]
Statistical Analysis 23: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 8, Day 56; Test type: Superiority; p = 0.0259, ANCOVA; Adjusted Difference = 0.42, 95% CI 2-sided [0.04 to 0.80]
Statistical Analysis 24: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 12, Day 84; Test type: Superiority; p = 0.9881, ANCOVA; Adjusted Difference = 0.06, 95% CI 2-sided [-0.34 to 0.46]
Statistical Analysis 25: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 12, Day 84; Test type: Superiority; p = 0.9891, ANCOVA; Adjusted Difference = 0.06, 95% CI 2-sided [-0.34 to 0.46]
Statistical Analysis 26: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 1, Day 7; Test type: Superiority; p = 0.0463, ANCOVA; Adjusted Difference = -0.29, 95% CI 2-sided [-0.57 to -0.00]
Statistical Analysis 27: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 2, Day 14; Test type: Superiority; p = 0.1867, ANCOVA; Adjusted Difference = -0.23, 95% CI 2-sided [-0.56 to 0.11]
Statistical Analysis 28: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0213, ANCOVA; Adjusted Difference = -0.44, 95% CI 2-sided [-0.81 to -0.07]
Statistical Analysis 29: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 8. Day 56; Test type: Superiority; p = 0.0003, ANCOVA; Adjusted Difference = -0.78, 95% CI 2-sided [-1.19 to -0.37]
Statistical Analysis 30: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0002, ANCOVA; Adjusted Difference = -0.82, 95% CI 2-sided [-1.24 to -0.40]

12. Secondary Outcome: Percentage of Participants With DAS Low Disease Activity
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. LDAS is defined as DAS28 ≤ 3.2
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Percentage of participants
  Week 1 Day 7 | 0.0 [0.00 to 0.00] | 0.9 [0.00 to 2.71] | 1.8 [0.00 to 4.31] | 0.0 [0.00 to 0.00] | 1.8 [0.00 to 4.28] | 2.1 [0.00 to 6.12] | 0.0 [0.00 to 0.00]
  Week 2 day 14 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 1.8 [0.00 to 4.31] | 0.9 [0.00 to 2.68] | 4.5 [0.65 to 8.36] | 2.1 [0.00 to 6.12] | 2.0 [0.00 to 5.88]
  Week 4 Day 28 | 0.0 [0.00 to 0.00] | 1.8 [0.00 to 4.35] | 6.4 [1.80 to 10.93] | 1.8 [0.00 to 4.31] | 11.7 [5.73 to 17.69] | 2.1 [0.00 to 6.12] | 0.0 [0.00 to 0.00]
  Week 8 Day 56 | 0.0 [0.00 to 0.00] | 8.3 [3.09 to 13.42] | 11.8 [5.79 to 17.85] | 3.6 [0.14 to 7.13] | 18.0 [10.87 to 25.17] | 2.1 [0.00 to 6.12] | 2.0 [0.00 to 5.88]
  Week 12 Day 84 | 7.5 [0.00 to 15.66] | 19.3 [11.86 to 26.67] | 14.5 [7.96 to 21.13] | 3.6 [0.14 to 7.13] | 17.1 [10.11 to 24.12] | 14.6 [4.60 to 24.57] | 4.0 [0.00 to 9.43]
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.06 to 6.06]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.5976, Cochran-Mantel-Haenszel; Adjusted Difference = 0.91, 95% CI 2-sided [-2.48 to 4.30]
Statistical Analysis 3: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.3482, Cochran-Mantel-Haenszel; Adjusted Difference = 1.82, 95% CI 2-sided [-1.98 to 5.62]
Statistical Analysis 4: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.8979, Cochran-Mantel-Haenszel; Adjusted Difference = -0.40, 95% CI 2-sided [-6.51 to 5.71]
Statistical Analysis 5: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.5976, Cochran-Mantel-Haenszel; Adjusted Difference = -0.91, 95% CI 2-sided [-4.30 to 2.48]
Statistical Analysis 6: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.6546, Cochran-Mantel-Haenszel; Adjusted Difference = 0.91, 95% CI 2-sided [-3.07 to 4.89]
Statistical Analysis 7: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4 Day 28; Test type: Superiority; p = 0.7988, Cochran-Mantel-Haenszel; Adjusted Difference = -0.80, 95% CI 2-sided [-6.95 to 5.35]
Statistical Analysis 8: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4 Day 28; Test type: Superiority; p = 0.9975, Cochran-Mantel-Haenszel; Adjusted Difference = 0.01, 95% CI 2-sided [-4.35 to 4.36]
Statistical Analysis 9: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.1185, Cochran-Mantel-Haenszel; Adjusted Difference = 4.55, 95% CI 2-sided [-1.16 to 10.25]
Statistical Analysis 10: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.4765, Cochran-Mantel-Haenszel; Adjusted Difference = -2.40, 95% CI 2-sided [-9.01 to 4.21]
Statistical Analysis 11: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.1655, Cochran-Mantel-Haenszel; Adjusted Difference = 4.61, 95% CI 2-sided [-1.90 to 11.12]
Statistical Analysis 12: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.0234, Cochran-Mantel-Haenszel; Adjusted Difference = 8.18, 95% CI 2-sided [1.11 to 15.26]
Statistical Analysis 13: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.5490, Cochran-Mantel-Haenszel; Adjusted Difference = 3.20, 95% CI 2-sided [-7.27 to 13.67]
Statistical Analysis 14: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Mean Difference (Net) = 15.62, 95% CI 2-sided [7.22 to 24.03]
Statistical Analysis 15: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0044, Cochran-Mantel-Haenszel; Adjusted Difference = 10.91, 95% CI 2-sided [3.39 to 18.43]
Statistical Analysis 16: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 1, Day 7; Test type: Superiority; p = 0.6588, Cochran-Mantel-Haenszel; Adjusted Difference = 2.05, 95% CI 2-sided [-7.07 to 11.18]
Statistical Analysis 17: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 2, Day 14; Test type: Superiority; p = 0.8853, Cochran-Mantel-Haenszel; Adjusted Difference = 0.68, 95% CI 2-sided [-8.62 to 9.99]
Statistical Analysis 18: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 4, Day 28; Test type: Superiority; p = 0.6564, Cochran-Mantel-Haenszel; Adjusted Difference = 2.05, 95% CI 2-sided [-7.00 to 11.11]
Statistical Analysis 19: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 8, Day 56; Test type: Superiority; p = 0.8853, Cochran-Mantel-Haenszel; Adjusted Difference = 0.68, 95% CI 2-sided [-8.62 to 9.99]
Statistical Analysis 20: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0584, Cochran-Mantel-Haenszel; Adjusted Difference = 11.64, 95% CI 2-sided [-0.41 to 23.70]

13. Secondary Outcome: Percentage of Participants With DAS Remission
Description: as for outcome 8
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Percentage of participants
  Week 1 Day 7 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 2.1 [0.00 to 6.12] | 0.0 [0.00 to 0.00]
  Week 2 Day 14 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.9 [0.00 to 2.68] | 0.0 [0.00 to 0.00] | 0.9 [0.00 to 2.66] | 0.00 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Week 4 Day 28 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 1.8 [0.00 to 4.31] | 0.9 [0.00 to 2.68] | 4.5 [0.65 to 8.36] | 0.00 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Week 8 Day 56 | 0.0 [0.00 to 0.00] | 3.7 [0.14 to 7.20] | 4.5 [0.65 to 8.44] | 1.8 [0.00 to 4.31] | 9.0 [3.68 to 14.34] | 0.00 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Week 12 Day 84 | 2.5 [0.00 to 7.34] | 7.3 [2.44 to 12.24] | 8.2 [3.06 to 13.30] | 3.6 [0.14 to 7.13] | 9.0 [3.68 to 14.34] | 4.2 [0.00 to 9.82] | 4.0 [0.00 to 9.43]
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.06 to 6.06]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-2.92 to 2.92]
Statistical Analysis 3: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-2.91 to 2.91]
Statistical Analysis 4: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.06 to 6.06]
Statistical Analysis 5: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-2.92 to 2.92]
Statistical Analysis 6: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.5976, Cochran-Mantel-Haenszel; Adjusted Difference = 0.91, 95% CI 2-sided [-2.47 to 4.28]
Statistical Analysis 7: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.8979, Cochran-Mantel-Haenszel; Adjusted Difference = -0.40, 95% CI 2-sided [-6.51 to 5.71]
Statistical Analysis 8: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4 Day 28; Test type: Superiority; p = 0.5976, Cochran-Mantel-Haenszel; Adjusted Difference = -0.91, 95% CI 2-sided [-4.30 to 2.48]
Statistical Analysis 9: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.6669, Cochran-Mantel-Haenszel; Adjusted Difference = 0.91, 95% CI 2-sided [-3.23 to 5.05]
Statistical Analysis 10: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.6309, Cochran-Mantel-Haenszel; Adjusted Difference = -1.60, 95% CI 2-sided [-8.13 to 4.93]
Statistical Analysis 11: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.4473, Cochran-Mantel-Haenszel; Adjusted Difference = 1.83, 95% CI 2-sided [-2.90 to 6.56]
Statistical Analysis 12: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.3021, Cochran-Mantel-Haenszel; Adjusted Difference = 2.73, 95% CI 2-sided [-2.45 to 7.91]
Statistical Analysis 13: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.7134, Cochran-Mantel-Haenszel; Adjusted Difference = -1.60, 95% CI 2-sided [-10.14 to 6.94]
Statistical Analysis 14: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.2635, Cochran-Mantel-Haenszel; Adjusted Difference = 3.70, 95% CI 2-sided [-2.79 to 10.19]
Statistical Analysis 15: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.1749, Cochran-Mantel-Haenszel; Adjusted Difference = 4.55, 95% CI 2-sided [-2.02 to 11.11]
Statistical Analysis 16: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 1, Day 7; Test type: Superiority; p = 0.6588, Cochran-Mantel-Haenszel; Adjusted Difference = 2.05, 95% CI 2-sided [-7.07 to 11.18]
Statistical Analysis 17: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 2 Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-8.31 to 8.31]
Statistical Analysis 18: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 4, Day 28; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-8.31 to 8.31]
Statistical Analysis 19: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 8, Day 56; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-8.31 to 8.31]
Statistical Analysis 20: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 12, Day 84; Test type: Superiority; p = 0.7848, Cochran-Mantel-Haenszel; Adjusted Difference = 1.37, 95% CI 2-sided [-8.46 to 11.20]

14. Secondary Outcome: Percentage of Participants Meeting the Boolean-based Remission Criteria
Description: Boolean Remission is defined as Tender joint count less than 1, Swollen joint count less than 1, CRP less than 1 mg/dL, patient global assessment less than 1 (on 0 to 10 VAS scale).
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Percentage of participants
  Week 1 Day 7: number analyzed (Participants) | 38 | 107 | 108 | 110 | 107 | 47 | 47
  Week 1 Day 7 | 0.0 [0.00 to 0.00] | 0.9 [0.00 to 2.76] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Week 2 Day 14: number analyzed (Participants) | 39 | 107 | 109 | 110 | 109 | 48 | 49
  Week 2 Day 14 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Week 4 Day 28: number analyzed (Participants) | 38 | 105 | 107 | 108 | 109 | 47 | 48
  Week 4 Day 28 | 0.0 [0.00 to 0.00] | 1.0 [0.00 to 2.81] | 0.0 [0.00 to 0.00] | 0.9 [0.00 to 2.73] | 2.8 [0.00 to 5.82] | 2.1 [0.00 to 6.25] | 0.0 [0.00 to 0.00]
  Week 8 Day 56: number analyzed (Participants) | 37 | 101 | 104 | 103 | 109 | 47 | 45
  Week 8 Day 56 | 0.0 [0.00 to 0.00] | 2.0 [0.00 to 4.70] | 1.90 [0.00 to 4.56] | 1.0 [0.00 to 2.86] | 3.7 [0.14 to 7.20] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Week 12 Day 84: number analyzed (Participants) | 37 | 98 | 97 | 102 | 108 | 47 | 45
  Week 12 Day 84 | 0.0 [0.00 to 0.00] | 2.0 [0.00 to 4.84] | 4.1 [0.17 to 8.08] | 1.0 [0.00 to 2.89] | 6.5 [1.84 to 11.12] | 8.5 [0.53 to 16.49] | 0.0 [0.00 to 6.53]
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.28 to 6.28]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.5941, Cochran-Mantel-Haenszel; Adjusted Difference = 0.93, 95% CI 2-sided [-2.50 to 4.37]
Statistical Analysis 3: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-2.93 to 2.93]
Statistical Analysis 4: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.17 to 6.17]
Statistical Analysis 5: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-2.95 to 2.95]
Statistical Analysis 6: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-2.92 to 2.92]
Statistical Analysis 7: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.8929, Cochran-Mantel-Haenszel; Adjusted Difference = -0.43, 95% CI 2-sided [-6.62 to 5.77]
Statistical Analysis 8: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.9424, Cochran-Mantel-Haenszel; Adjusted Difference = -0.13, 95% CI 2-sided [-3.78 to 3.51]
Statistical Analysis 9: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.5927, Cochran-Mantel-Haenszel; Adjusted Difference = -0.94, 95% CI 2-sided [-4.40 to 2.51]
Statistical Analysis 10: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.8788, Cochran-Mantel-Haenszel; Adjusted Difference = -0.46, 95% CI 2-sided [-6.31 to 5.40]
Statistical Analysis 11: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8 Day 56; Test type: Superiority; p = 0.6876, Cochran-Mantel-Haenszel; Adjusted Difference = 0.87, 95% CI 2-sided [-3.36 to 5.09]
Statistical Analysis 12: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.6656, Cochran-Mantel-Haenszel; Adjusted Difference = 0.97, 95% CI 2-sided [-3.42 to 5.35]
Statistical Analysis 13: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12 Day 84; Test type: Superiority; p = 0.8787, Cochran-Mantel-Haenszel; Adjusted Difference = -0.46, 95% CI 2-sided [-6.34 to 5.42]
Statistical Analysis 14: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.7101, Cochran-Mantel-Haenszel; Adjusted Difference = 0.74, 95% CI 2-sided [-3.17 to 4.66]
Statistical Analysis 15: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.2425, Cochran-Mantel-Haenszel; Adjusted Difference = 3.20, 95% CI 2-sided [-2.16 to 8.55]
Statistical Analysis 16: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 1, Day 7; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-8.68 to 8.68]
Statistical Analysis 17: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 2 Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-8.39 to 8.39]
Statistical Analysis 18: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 4, Day 28; Test type: Superiority; p = 0.6658, Cochran-Mantel-Haenszel; Adjusted Difference = 2.03, 95% CI 2-sided [-7.17 to 11.22]
Statistical Analysis 19: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 8, Day 56; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-8.77 to 8.77]
Statistical Analysis 20: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 12, Day 84; Test type: Superiority; p = 0.2457, Cochran-Mantel-Haenszel; Adjusted Difference = 6.57, 95% CI 2-sided [-4.52 to 17.66]

15. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI)
Description: CDAI was derived as the sum of the following: tender joint count (TJC), swollen joint count (SJC), participant global assessment (PGA) of disease activity, and physician assessment of disease activity. TJC and SJC were taken as the number of tender and swollen joints, respectively, out of 28 assessed joints. PGA and physician assessment of disease activity were scored 0-100 millimeters (mm) and rounded to the nearest centimeter (cm) on a visual analog scale (VAS), where higher scores indicate greater perceived disease activity. The total CDAI score range was 0-76, where higher scores indicate increased disease activity. Change from baseline at a particular time point was calculated among patients with data available at both baseline and the time point of interest. Negative values indicate improvement/reduction in RA disease activity.
Time Frame: Baseline, Days 7, 14, 28, 56 and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale
  Week 1 Day 7: number analyzed (Participants) | 38 | 105 | 103 | 104 | 104 | 47 | 45
  Week 1 Day 7 | -5.45 (7.69) | -6.70 (8.26) | -7.40 (9.97) | -4.71 (12.91) | -9.64 (8.93) | -8.61 (10.67) | -5.26 (9.79)
  Week 2 Day 14: number analyzed (Participants) | 38 | 103 | 106 | 105 | 107 | 48 | 47
  Week 2 Day 14 | -6.85 (11.10) | -10.33 (10.45) | -11.33 (10.47) | -7.44 (13.39) | -13.44 (10.52) | -9.64 (12.17) | -7.70 (10.64)
  Week 4 Day 28: number analyzed (Participants) | 37 | 100 | 100 | 99 | 105 | 47 | 48
  Week 4 Day 28 | -10.36 (10.88) | -13.84 (12.11) | -13.78 (11.46) | -9.43 (14.77) | -17.74 (10.84) | -11.83 (11.08) | -7.49 (11.46)
  Week 8 Day 56: number analyzed (Participants) | 37 | 100 | 100 | 99 | 105 | 47 | 44
  Week 8 Day 56 | -14.76 (10.04) | -18.61 (13.48) | -18.10 (12.99) | -15.49 (15.74) | -21.36 (11.69) | -17.38 (12.39) | -7.57 (10.51)
  Week 12 Day 84: number analyzed (Participants) | 36 | 95 | 94 | 99 | 105 | 47 | 44
  Week 12 Day 84 | -16.99 (11.21) | -22.05 (12.19) | -22.10 (11.83) | -17.02 (16.24) | -22.22 (11.76) | -20.42 (13.20) | -12.23 (12.06)
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.4960, Cochran-Mantel-Haenszel; Adjusted Difference = -2.36, 95% CI 2-sided [-6.73 to 2.02]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.2736, Cochran-Mantel-Haenszel; Adjusted Difference = -2.18, 95% CI 2-sided [-5.34 to 0.98]
Statistical Analysis 3: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.0608, Cochran-Mantel-Haenszel; Adjusted Difference = -3.08, 95% CI 2-sided [-6.26 to 0.10]
Statistical Analysis 4: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.9237, Cochran-Mantel-Haenszel; Adjusted Difference = -1.25, 95% CI 2-sided [-6.02 to 3.52]
Statistical Analysis 5: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.0893, Cochran-Mantel-Haenszel; Adjusted Difference = -3.14, 95% CI 2-sided [-6.60 to 0.33]
Statistical Analysis 6: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 0.0138, Cochran-Mantel-Haenszel; Adjusted Difference = -4.07, 95% CI 2-sided [-7.51 to -0.63]
Statistical Analysis 7: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.3358, Cochran-Mantel-Haenszel; Adjusted Difference = -3.22, 95% CI 2-sided [-8.24 to 1.80]
Statistical Analysis 8: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0078, Cochran-Mantel-Haenszel; Adjusted Difference = -4.57, 95% CI 2-sided [-8.20 to -0.94]
Statistical Analysis 9: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0059, Cochran-Mantel-Haenszel; Adjusted Difference = -4.68, 95% CI 2-sided [-8.30 to -1.06]
Statistical Analysis 10: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.6503, Cochran-Mantel-Haenszel; Adjusted Difference = -2.29, 95% CI 2-sided [-7.39 to 2.80]
Statistical Analysis 11: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.1282, Cochran-Mantel-Haenszel; Adjusted Difference = -3.12, 95% CI 2-sided [-6.84 to 0.59]
Statistical Analysis 12: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.1675, Cochran-Mantel-Haenszel; Adjusted Difference = -2.94, 95% CI 2-sided [-6.65 to 0.78]
Statistical Analysis 13: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.4220, Cochran-Mantel-Haenszel; Adjusted Difference = -2.94, 95% CI 2-sided [-7.96 to 2.09]
Statistical Analysis 14: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0027, Cochran-Mantel-Haenszel; Adjusted Difference = -5.10, 95% CI 2-sided [-8.77 to -1.42]
Statistical Analysis 15: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0011, Cochran-Mantel-Haenszel; Adjusted Difference = -5.47, 95% CI 2-sided [-9.15 to -1.78]
Statistical Analysis 16: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 1, Day 7; Test type: Superiority; p = 0.0455, Cochran-Mantel-Haenszel; Adjusted Difference = 3.21, 95% CI 2-sided [0.05 to 6.37]
Statistical Analysis 17: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 1, Day 7; Test type: Superiority; p = 0.2309, Cochran-Mantel-Haenszel; Adjusted Difference = 2.31, 95% CI 2-sided [-0.87 to 5.48]
Statistical Analysis 18: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 2, Day 14; Test type: Superiority; p = 0.0698, Cochran-Mantel-Haenszel; Adjusted Difference = 3.27, 95% CI 2-sided [-0.18 to 6.72]
Statistical Analysis 19: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 2, Day 14; Test type: Superiority; p = 0.2851, Cochran-Mantel-Haenszel; Adjusted Difference = 2.33, 95% CI 2-sided [-1.09 to 5.76]
Statistical Analysis 20: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 4, Day 28; Test type: Superiority; p = 0.0131, Cochran-Mantel-Haenszel; Adjusted Difference = 4.29, 95% CI 2-sided [0.69 to 7.90]
Statistical Analysis 21: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 4, Day 28; Test type: Superiority; p = 0.0161, Cochran-Mantel-Haenszel; Adjusted Difference = 4.18, 95% CI 2-sided [0.59 to 7.78]
Statistical Analysis 22: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 8, Day 56; Test type: Superiority; p = 0.0360, Cochran-Mantel-Haenszel; Adjusted Difference = 3.85, 95% CI 2-sided [0.18 to 7.51]
Statistical Analysis 23: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 8, Day 56; Test type: Superiority; p = 0.0252, Cochran-Mantel-Haenszel; Adjusted Difference = 4.04, 95% CI 2-sided [0.37 to 7.70]
Statistical Analysis 24: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 12, Day 84; Test type: Superiority; p = 0.9032, Cochran-Mantel-Haenszel; Adjusted Difference = 1.03, 95% CI 2-sided [-2.59 to 4.66]
Statistical Analysis 25: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 12, Day 84; Test type: Superiority; p = 0.9791, Cochran-Mantel-Haenszel; Adjusted Difference = 0.66, 95% CI 2-sided [-2.97 to 4.30]
Statistical Analysis 26: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 1, Day 7; Test type: Superiority; p = 0.0927, Cochran-Mantel-Haenszel; Adjusted Difference = -3.22, 95% CI 2-sided [-6.98 to 0.54]
Statistical Analysis 27: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 2, Day 14; Test type: Superiority; p = 0.3202, Cochran-Mantel-Haenszel; Adjusted Difference = -2.12, 95% CI 2-sided [-6.33 to 2.09]
Statistical Analysis 28: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0476, Cochran-Mantel-Haenszel; Adjusted Difference = -4.20, 95% CI 2-sided [-8.36 to -0.04]
Statistical Analysis 29: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 8, Day 54; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Difference = -9.93, 95% CI 2-sided [-14.31 to -5.55]
Statistical Analysis 30: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Adjusted Difference = -8.23, 95% CI 2-sided [-12.56 to -3.90]

16. Secondary Outcome: Percentage of Participants Meeting the CDAI-based Remission Criteria
Description: Clinical Disease Activity Index is defined as CDAI= : SJC(28) + TJC(28) + PGA + MDG where TJC and SJC are the tender and swollen joint counts from 28 joints, PGA is the patient's global assessment of disease activity (on a 0-10 scale) and MDG is physician global assessment of disease activity (on a 0-10 scale). The cutoff value for CDAI remission is <=2.8.
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Percentage of participants
  Week 1 Day 7 | 0.0 [0.00 to 0.00] | 0.9 [0.00 to 2.71] | 0.9 [0.00 to 2.68] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Week 2 Day 14 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 1.8 [0.00 to 4.28] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Week 4 Day 28 | 0.0 [0.00 to 0.00] | 0.9 [0.00 to 2.71] | 0.9 [0.00 to 2.68] | 0.0 [0.00 to 0.00] | 4.5 [0.65 to 8.36] | 2.1 [0.00 to 6.12] | 0.0 [0.00 to 0.00]
  Week 8 Day 56 | 0.0 [0.00 to 0.00] | 2.8 [0.00 to 5.82] | 5.5 [1.21 to 9.70] | 0.00 [0.00 to 0.00] | 7.2 [2.40 to 12.02] | 4.2 [0.00 to 9.82] | 0.0 [0.00 to 0.00]
  Week 12 Day 84 | 0.0 [0.00 to 0.00] | 5.5 [1.22 to 9.79] | 6.4 [1.80 to 10.93] | 0.9 [0.00 to 2.68] | 9.9 [4.35 to 15.47] | 6.3 [0.00 to 13.10] | 6.0 [0.00 to 12.58]
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.06 to 6.06]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.5976, Cochran-Mantel-Haenszel; Adjusted Difference = 0.91, 95% CI 2-sided [-2.48 to 4.30]
Statistical Analysis 3: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.5976, Cochran-Mantel-Haenszel; Adjusted Difference = 0.91, 95% CI 2-sided [-2.47 to 4.28]
Statistical Analysis 4: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.06 to 6.06]
Statistical Analysis 5: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-2.92 to 2.92]
Statistical Analysis 6: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-2.91 to 2.91]
Statistical Analysis 7: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.06 to 6.06]
Statistical Analysis 8: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.5726, Cochran-Mantel-Haenszel; Adjusted Difference = 0.91, 95% CI 2-sided [-2.26 to 4.09]
Statistical Analysis 9: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.5976, Cochran-Mantel-Haenszel; Adjusted Difference = 0.91, 95% CI 2-sided [-2.47 to 4.28]
Statistical Analysis 10: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.06 to 6.06]
Statistical Analysis 11: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.1446, Cochran-Mantel-Haenszel; Adjusted Difference = 2.74, 95% CI 2-sided [-0.94 to 6.42]
Statistical Analysis 12: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.0286, Cochran-Mantel-Haenszel; Adjusted Difference = 5.45, 95% CI 2-sided [0.57 to 10.34]
Statistical Analysis 13: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.8979, Cochran-Mantel-Haenszel; Adjusted Difference = -0.40, 95% CI 2-sided [-6.51 to 5.71]
Statistical Analysis 14: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0708, Cochran-Mantel-Haenszel; Adjusted Difference = 4.57, 95% CI 2-sided [-0.39 to 9.52]
Statistical Analysis 15: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0478, Cochran-Mantel-Haenszel; Adjusted Difference = 5.45, 95% CI 2-sided [0.05 to 10.86]
Statistical Analysis 16: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 1, Day 7; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-8.31 to 8.31]
Statistical Analysis 17: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-8.31 to 8.31]
Statistical Analysis 18: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 4, Day 28; Test type: Superiority; p = 0.6564, Cochran-Mantel-Haenszel; Adjusted Difference = 2.05, 95% CI 2-sided [-7.00 to 11.11]
Statistical Analysis 19: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 8, Day 56; Test type: Superiority; p = 0.3838, Cochran-Mantel-Haenszel; Adjusted Difference = 4.11, 95% CI 2-sided [-5.14 to 13.36]
Statistical Analysis 20: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 12, Day 84; Test type: Superiority; p = 0.9009, Cochran-Mantel-Haenszel; Adjusted Difference = 0.68, 95% CI 2-sided [-10.10 to 11.47]

17. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI)
Description: Simplified Disease Activity Index (SDAI) is the numerical sum of five outcome parameters: TJC and SJC (based on a 28-joint assessment), PtGA and PhGA (based on 0-10 cm VAS, where 0 = no disease activity and 10 = worst disease activity), and CRP. SDAI total score ranges from 0 (no disease activity) to 86 (maximal disease activity), where higher scores represents higher disease activity. The SDAI =< 3.3 indicates disease remission, > 3.4 to 11 indicates low disease activity, > 11 to 26 indicates moderate disease activity, and > 26 indicates high disease activity
Time Frame: Baseline, Days 7, 14, 28, 56 and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale
  Week 1 Day 7: number analyzed (Participants) | 37 | 104 | 102 | 103 | 104 | 47 | 45
  Week 1 Day 7 | -5.36 (7.86) | -6.48 (8.87) | -6.99 (10.49) | -4.75 (13.25) | -10.86 (9.33) | -8.73 (11.21) | -5.37 (9.49)
  Week 2 Day 14: number analyzed (Participants) | 37 | 103 | 105 | 105 | 107 | 48 | 46
  Week 2 Day 14 | -6.50 (10.54) | -10.46 (10.97) | -11.44 (10.85) | -7.54 (13.74) | -14.39 (10.99) | -9.84 (12.29) | -8.13 (11.01)
  Week 4 Day 28: number analyzed (Participants) | 36 | 101 | 103 | 99 | 105 | 47 | 48
  Week 4 Day 28 | -10.53 (11.03) | -14.47 (12.41) | -14.21 (12.20) | -8.92 (15.17) | -18.87 (11.20) | -12.13 (11.13) | -7.74 (12.02)
  Week 8 Day 56: number analyzed (Participants) | 36 | 99 | 100 | 97 | 103 | 47 | 44
  Week 8 Day 56 | -15.25 (10.41) | -18.95 (13.80) | -18.97 (13.91) | -15.74 (16.18) | -22.62 (11.97) | -18.57 (12.80) | -7.82 (11.20)
  Week 12 Day 84: number analyzed (Participants) | 36 | 94 | 94 | 99 | 103 | 47 | 43
  Week 12 Day 84 | -17.54 (11.36) | -22.89 (12.52) | -23.24 (12.50) | -17.47 (16.70) | -23.33 (11.97) | -21.97 (13.78) | -12.92 (12.61)
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.5455, Cochran-Mantel-Haenszel; Adjusted Difference = -2.36, 95% CI 2-sided [-7.00 to 2.27]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.4114, Cochran-Mantel-Haenszel; Adjusted Difference = -1.97, 95% CI 2-sided [-5.30 to 1.36]
Statistical Analysis 3: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.1739, Cochran-Mantel-Haenszel; Adjusted Difference = -2.62, 95% CI 2-sided [-5.97 to 0.72]
Statistical Analysis 4: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Week 14; Test type: Superiority; p = 0.9761, Cochran-Mantel-Haenszel; Adjusted Difference = -0.94, 95% CI 2-sided [-5.93 to 4.06]
Statistical Analysis 5: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Week 14; Test type: Superiority; p = 0.0998, Cochran-Mantel-Haenszel; Adjusted Difference = -3.18, 95% CI 2-sided [-6.78 to 0.41]
Statistical Analysis 6: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Week 14; Test type: Superiority; p = 0.0239, Cochran-Mantel-Haenszel; Adjusted Difference = -3.97, 95% CI 2-sided [-7.54 to -0.39]
Statistical Analysis 7: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.2018, Cochran-Mantel-Haenszel; Adjusted Difference = -3.98, 95% CI 2-sided [-9.25 to 1.30]
Statistical Analysis 8: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0011, Cochran-Mantel-Haenszel; Adjusted Difference = -5.67, 95% CI 2-sided [-9.48 to -1.87]
Statistical Analysis 9: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0026, Cochran-Mantel-Haenszel; Adjusted Difference = -5.27, 95% CI 2-sided [-9.06 to -1.48]
Statistical Analysis 10: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.6336, Cochran-Mantel-Haenszel; Adjusted Difference = -2.47, 95% CI 2-sided [-7.84 to 2.90]
Statistical Analysis 11: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.0950, Cochran-Mantel-Haenszel; Adjusted Difference = -3.49, 95% CI 2-sided [-7.38 to 0.41]
Statistical Analysis 12: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.1451, Cochran-Mantel-Haenszel; Adjusted Difference = -3.18, 95% CI 2-sided [-7.06 to 0.71]
Statistical Analysis 13: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.3434, Cochran-Mantel-Haenszel; Adjusted Difference = -3.28, 95% CI 2-sided [-8.43 to 1.87]
Statistical Analysis 14: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0016, Cochran-Mantel-Haenszel; Adjusted Difference = -5.45, 95% CI 2-sided [-9.23 to -1.68]
Statistical Analysis 15: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel; Adjusted Difference = -5.88, 95% CI 2-sided [-9.65 to -2.10]
Statistical Analysis 16: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 1, Day 7; Test type: Superiority; p = 0.0025, Cochran-Mantel-Haenszel; Adjusted Difference = 4.64, 95% CI 2-sided [1.31 to 7.96]
Statistical Analysis 17: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 1, Day 7; Test type: Superiority; p = 0.0129, Cochran-Mantel-Haenszel; Adjusted Difference = 3.98, 95% CI 2-sided [0.64 to 7.32]
Statistical Analysis 18: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 2, Day 14; Test type: Superiority; p = 0.0206, Cochran-Mantel-Haenszel; Adjusted Difference = 4.04, 95% CI 2-sided [0.46 to 7.62]
Statistical Analysis 19: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 2, Day 14; Test type: Superiority; p = 0.0841, Cochran-Mantel-Haenszel; Adjusted Difference = 3.26, 95% CI 2-sided [-0.30 to 6.82]
Statistical Analysis 20: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 4, Day 28; Test type: Superiority; p = 0.0088, Cochran-Mantel-Haenszel; Adjusted Difference = 4.67, 95% CI 2-sided [0.91 to 8.42]
Statistical Analysis 21: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 4, Day 28; Test type: Superiority; p = 0.0034, Cochran-Mantel-Haenszel; Adjusted Difference = 5.07, 95% CI 2-sided [1.34 to 8.81]
Statistical Analysis 22: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 8, Day 56; Test type: Superiority; p = 0.0138, Cochran-Mantel-Haenszel; Adjusted Difference = 4.55, 95% CI 2-sided [0.71 to 8.39]
Statistical Analysis 23: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 8, Day 56; Test type: Superiority; p = 0.0073, Cochran-Mantel-Haenszel; Adjusted Difference = 4.85, 95% CI 2-sided [1.02 to 8.69]
Statistical Analysis 24: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 12, Day 84; Test type: Superiority; p = 0.8284, Cochran-Mantel-Haenszel; Adjusted Difference = 1.29, 95% CI 2-sided [-2.46 to 5.03]
Statistical Analysis 25: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab; Week 12, Day 84; Test type: Superiority; p = 0.9525, Cochran-Mantel-Haenszel; Adjusted Difference = 0.86, 95% CI 2-sided [-2.88 to 4.60]
Statistical Analysis 26: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 1, Day 7; Test type: Superiority; p = 0.0856, Cochran-Mantel-Haenszel; Adjusted Difference = -3.22, 95% CI 2-sided [-6.91 to 0.46]
Statistical Analysis 27: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 2, Day 14; Test type: Superiority; p = 0.3374, Cochran-Mantel-Haenszel; Adjusted Difference = -2.08, 95% CI 2-sided [-6.36 to 2.20]
Statistical Analysis 28: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 4, Day 28; Test type: Superiority; p = 0.0534, Cochran-Mantel-Haenszel; Adjusted Difference = -4.24, 95% CI 2-sided [-8.53 to 0.06]
Statistical Analysis 29: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 8, Day 56; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Difference = -10.8, 95% CI 2-sided [-15.33 to -6.32]
Statistical Analysis 30: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 12, Day 84; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Difference = -9.22, 95% CI 2-sided [-13.63 to -4.81]

18. Secondary Outcome: Percentage of Participants Meeting the SDAI-based Remission Criteria
Description: The SDAI was the numerical sum of five outcome parameter: SJC and TJC (based on a 28-joint assessment), PGA and MDG (based on 0-10 cm VAS, where 0 = no disease activity and 10 = worst disease activity), and CRP. The SDAI =< 3.3 indicates disease remission
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Percentage of participants
  Week 1 Day 7 | 0.00 [0.00 to 0.00] | 0.9 [0.00 to 2.71] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 2 Day 14 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 1.8 [0.00 to 4.28] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 4 Day 28 | 0.00 [0.00 to 0.00] | 0.9 [0.00 to 2.71] | 0.9 [0.00 to 2.68] | 0.00 [0.00 to 0.00] | 4.5 [0.65 to 8.36] | 2.1 [0.00 to 6.12] | 0.00 [0.00 to 0.00]
  Week 8 Day 56 | 0.00 [0.00 to 0.00] | 2.8 [0.00 to 5.82] | 3.6 [0.14 to 7.13] | 0.00 [0.00 to 0.00] | 6.3 [1.78 to 10.83] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Week 12 Day 84 | 0.00 [0.00 to 0.00] | 4.6 [0.66 to 8.51] | 6.4 [1.80 to 10.93] | 0.9 [0.00 to 2.68] | 9.0 [3.68 to 14.34] | 6.3 [0.00 to 13.10] | 6.0 [0.00 to 12.58]
Statistical Analysis 1: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.06 to 6.06]
Statistical Analysis 2: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 0.5976, Cochran-Mantel-Haenszel; Adjusted Difference = 0.91, 95% CI 2-sided [-2.48 to 4.30]
Statistical Analysis 3: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 1, Day 7; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-2.91 to 2.91]
Statistical Analysis 4: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.06 to 6.06]
Statistical Analysis 5: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-2.92 to 2.92]
Statistical Analysis 6: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-2.91 to 2.91]
Statistical Analysis 7: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.06 to 6.06]
Statistical Analysis 8: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.5726, Cochran-Mantel-Haenszel; Adjusted Difference = 0.91, 95% CI 2-sided [-2.26 to 4.09]
Statistical Analysis 9: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 4, Day 28; Test type: Superiority; p = 0.5976, Cochran-Mantel-Haenszel; Mean Difference (Net) = 0.91, 95% CI 2-sided [-2.47 to 4.28]
Statistical Analysis 10: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-6.06 to 6.06]
Statistical Analysis 11: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.1446, Cochran-Mantel-Haenszel; Adjusted Difference = 2.74, 95% CI 2-sided [-0.94 to 6.42]
Statistical Analysis 12: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 8, Day 56; Test type: Superiority; p = 0.1050, Cochran-Mantel-Haenszel; Adjusted Difference = 3.64, 95% CI 2-sided [-0.76 to 8.03]
Statistical Analysis 13: Comparison: Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.8979, Cochran-Mantel-Haenszel; Adjusted Difference = -0.40, 95% CI 2-sided [-6.51 to 5.71]
Statistical Analysis 14: Comparison: Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.1270, Cochran-Mantel-Haenszel; Adjusted Difference = 3.65, 95% CI 2-sided [-1.04 to 8.35]
Statistical Analysis 15: Comparison: Cohort 1: GDC-0853 High Dose + Adalimumab Placebo vs Cohort 1: GDC-0853 Placebo + Adalimumab Placebo; Week 12, Day 84; Test type: Superiority; p = 0.0501, Cochran-Mantel-Haenszel; Adjusted Difference = 5.45, 95% CI 2-sided [-0.00 to 10.91]
Statistical Analysis 16: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 1, Day 7; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-8.31 to 8.31]
Statistical Analysis 17: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 2, Day 14; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-8.31 to 8.31]
Statistical Analysis 18: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 4, Day 28; Test type: Superiority; p = 0.6564, Cochran-Mantel-Haenszel; Adjusted Difference = 2.05, 95% CI 2-sided [-7.00 to 11.11]
Statistical Analysis 19: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 8, Day 56; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel; Adjusted Difference = 0.00, 95% CI 2-sided [-8.31 to 8.31]
Statistical Analysis 20: Comparison: Cohort 2: GDC-0853 High Dose vs Cohort 2: GDC-0853 Placebo; Week 12, Day 84; Test type: Superiority; p = 0.9051, Cochran-Mantel-Haenszel; Adjusted Difference = 0.68, 95% CI 2-sided [-10.58 to 11.95]

19. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Version 2.0 (V2) Scores for Physical and Mental Components
Description: The 36-Item Short Form Health Survey (SF-36v2) is a questionnaire used to assess functional health and well-being and consists of eight domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health.
  The SF-36v2 is summarized into Physical Component Summary (PCS) and Mental Component Summary (MCS) scores. The PCS and MCS scores range from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A positive change from baseline indicates improvement.
Time Frame: Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Number on a scale
  Physical component score change: baseline-week 12: number analyzed (Participants) | 35 | 98 | 100 | 99 | 106 | 45 | 44
  Physical component score change: baseline-week 12 | 5.57 (5.98) | 5.71 (6.85) | 6.59 (7.54) | 3.54 (6.81) | 6.41 (6.43) | 5.35 (7.48) | 1.75 (6.39)
  Mental component score change: baseline-week 12: number analyzed (Participants) | 36 | 98 | 101 | 99 | 106 | 45 | 43
  Mental component score change: baseline-week 12 | 7.04 (9.32) | 4.89 (10.57) | 6.92 (12.06) | 4.29 (10.51) | 6.50 (10.79) | 5.76 (10.22) | 5.11 (10.10)

20. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score
Description: The FACIT-Fatigue Scale consists of 13 items designed to measure the degree of fatigue experienced by the patient in the previous 7 days. For each question, there are five possible responses: 0 (not at all), 1 (a little bit), 2 (somewhat), 3 (quite a bit), 4 (very much).
  A total fatigue score is calculated by summing all items, and possible total scores range from 0 (maximum fatigue) to 52 (no fatigue). A positive change from baseline indicates an improvement in the patient's fatigue (less fatigue).
Time Frame: Day 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale | 9.00 (10.57) | 8.21 (10.22) | 8.95 (10.04) | 7.08 (10.88) | 9.59 (9.02) | 8.85 (9.57) | 5.71 (9.24)

21. Secondary Outcome: Change From Baseline in Tender/Painful Joint Count (68 Joint Count)
Description: Tender Joint Count: a total of 68 joints will be assessed for tenderness. Each joint is assessed for the presence/absence of tenderness. 68 joints are assessed for tenderness and joints are classified as tender/not tender giving a total possible tender joint count score of 0 to 68. A negative change from Baseline indicated improvement.
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale
  Week 1 Day 7: number analyzed (Participants) | 38 | 107 | 108 | 110 | 107 | 47 | 47
  Week 1 Day 7 | -2.79 (7.25) | -4.12 (8.14) | -3.33 (9.27) | -3.81 (10.85) | -5.58 (9.41) | -6.57 (8.66) | -3.06 (11.01)
  Week 2 Day 19: number analyzed (Participants) | 39 | 108 | 110 | 110 | 109 | 48 | 50
  Week 2 Day 19 | -4.33 (12.31) | -6.36 (10.88) | -5.91 (9.38) | -5.78 (11.50) | -8.62 (10.46) | -6.08 (8.53) | -3.92 (10.77)
  Week 4 Day 28: number analyzed (Participants) | 39 | 108 | 110 | 110 | 109 | 48 | 50
  Week 4 Day 28 | -6.00 (8.89) | -7.90 (11.28) | -6.84 (9.53) | -7.55 (12.97) | -11.61 (11.43) | -7.79 (7.93) | -4.40 (12.37)
  Week 8 Day 56: number analyzed (Participants) | 39 | 109 | 110 | 110 | 109 | 48 | 50
  Week 8 Day 56 | -9.72 (8.20) | -11.57 (12.18) | -9.75 (10.93) | -10.75 (14.37) | -14.12 (11.33) | -11.65 (10.34) | -4.60 (12.41)
  Week 12 Day 84: number analyzed (Participants) | 39 | 109 | 110 | 110 | 109 | 48 | 50
  Week 12 Day 84 | -10.33 (9.40) | -12.72 (12.05) | -11.49 (11.15) | -10.55 (14.37) | -15.49 (12.31) | -13.73 (12.81) | -7.14 (13.32)

22. Secondary Outcome: Change From Baseline in Swollen Joint Count (66 Joint Count)
Description: Swollen Joint Count: a total of 66 joints will be assessed for swelling. Each joint is assessed for the presence/absence of swelling. 66 joints were assessed for swelling and joints are classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66. A negative change from Baseline indicated improvement.
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale
  Week 1 Day 7: number analyzed (Participants) | 38 | 107 | 108 | 110 | 107 | 47 | 47
  Week 1 Day 7 | -1.84 (5.19) | -2.89 (5.01) | -3.45 (6.02) | -3.35 (9.38) | -3.94 (5.33) | -3.45 (4.90) | -1.49 (4.49)
  Week 2 Day 14: number analyzed (Participants) | 39 | 108 | 110 | 110 | 109 | 48 | 50
  Week 2 Day 14 | -3.95 (6.44) | -4.78 (5.99) | -5.06 (5.14) | -4.23 (9.88) | -6.26 (5.98) | -3.29 (5.69) | -2.96 (6.27)
  Week 4 Day 28: number analyzed (Participants) | 39 | 108 | 110 | 110 | 109 | 48 | 50
  Week 4 Day 28 | -4.38 (4.55) | -6.33 (7.98) | -5.95 (6.09) | -5.47 (9.26) | -8.50 (6.39) | -4.21 (6.39) | -3.46 (5.62)
  Week 8 Day 56: number analyzed (Participants) | 39 | 109 | 110 | 110 | 109 | 48 | 50
  Week 8 Day 56 | -6.54 (5.78) | -8.06 (8.13) | -7.72 (7.44) | -7.41 (10.82) | -9.60 (6.94) | -6.81 (6.16) | -3.02 (7.76)
  Week 12 Day 84: number analyzed (Participants) | 39 | 109 | 110 | 110 | 109 | 48 | 50
  Week 12 Day 84 | -7.36 (5.88) | -8.89 (8.23) | -8.48 (7.01) | -8.26 (11.48) | -9.94 (6.91) | -7.65 (6.75) | -4.86 (5.84)

23. Secondary Outcome: Change From Baseline in Patient Assessment Score of Arthritis Pain
Description: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale
  Week 1 Day 7: number analyzed (Participants) | 38 | 104 | 102 | 104 | 104 | 47 | 45
  Week 1 Day 7 | -9.00 (18.66) | -9.20 (20.56) | -11.18 (21.64) | -4.12 (22.43) | -15.75 (18.71) | -11.94 (21.25) | -2.76 (18.24)
  Week 2 Day 14: number analyzed (Participants) | 38 | 104 | 106 | 105 | 107 | 48 | 46
  Week 2 Day 14 | -6.08 (21.64) | -12.16 (20.09) | -17.08 (23.46) | -8.22 (25.72) | -18.13 (17.71) | -15.08 (21.87) | -4.72 (17.64)
  Week 4 Day 28: number analyzed (Participants) | 37 | 102 | 104 | 103 | 107 | 47 | 48
  Week 4 Day 28 | -13.41 (16.79) | -15.75 (21.97) | -18.63 (24.87) | -10.08 (27.16) | -20.21 (21.97) | -16.64 (27.86) | -7.54 (23.80)
  Week 8 Day 56: number analyzed (Participants) | 37 | 100 | 100 | 99 | 105 | 47 | 45
  Week 8 Day 56 | -18.38 (19.35) | -23.21 (22.10) | -25.95 (27.50) | -16.37 (27.65) | -24.70 (22.23) | -21.21 (27.13) | -7.13 (25.73)
  Week 12 Day 84: number analyzed (Participants) | 36 | 95 | 95 | 99 | 105 | 47 | 44
  Week 12 Day 84 | -23.14 (21.14) | -26.48 (23.30) | -30.63 (28.49) | -17.88 (29.42) | -26.30 (23.87) | -26.49 (27.65) | -13.98 (25.32)

24. Secondary Outcome: Change From Baseline in Patient Global Assessment Score of Arthritis Pain
Description: Participant-assessed arthritis pain was scored on a 100-mm VAS, where the distance from 0 mm represented the participant's self evaluation of arthritis pain (0 mm=none; 100 mm=very severe). Change from baseline at a particular time point was calculated among patients with data available at both baseline and the time point of interest, where negative change indicated a decrease in participant-assessed arthritis pain.
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale
  Week 1 Day 7: number analyzed (Participants) | 38 | 105 | 103 | 104 | 104 | 47 | 45
  Week 1 Day 7 | -9.00 (15.88) | -10.30 (20.82) | -11.82 (22.52) | -3.07 (20.83) | -18.33 (20.81) | -13.15 (22.17) | -4.96 (19.18)
  Week 2 Day 14: number analyzed (Participants) | 38 | 103 | 106 | 105 | 107 | 48 | 47
  Week 2 Day 14 | -5.50 (20.98) | -13.70 (19.63) | -14.84 (24.08) | -5.39 (26.13) | -18.94 (22.33) | -15.46 (21.67) | -8.64 (19.43)
  Week 4 Day 28: number analyzed (Participants) | 37 | 103 | 104 | 102 | 106 | 47 | 48
  Week 4 Day 28 | -12.11 (16.68) | 16.10 (23.48) | -17.75 (22.73) | -6.36 (25.99) | -21.78 (25.53) | -18.26 (27.53) | -10.96 (21.54)
  Week 8 Day 56: number analyzed (Participants) | 37 | 100 | 100 | 99 | 105 | 47 | 45
  Week 8 Day 56 | -19.19 (16.88) | -24.06 (24.99) | -22.59 (26.81) | -14.19 (29.80) | -26.77 (25.69) | -21.17 (25.98) | -11.82 (21.66)
  Week 12 Day 84: number analyzed (Participants) | 36 | 95 | 95 | 99 | 106 | 47 | 44
  Week 12 Day 84 | -23.33 (22.03) | -26.67 (26.89) | -27.33 (27.33) | -16.87 (28.68) | -26.24 (27.02) | -25.55 (27.52) | -13.80 (22.17)

25. Secondary Outcome: Change From Baseline in Physician's Global Assessment Score of Arthritis
Description: Physician's assessment of participant's disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the physician's assessment of the participant's disease activity (0 mm=very good; 100 mm=very poor). Change from baseline at a particular time point was calculated among patients with data available at both baseline and the time point of interest, where negative change from baseline indicated an improvement in physician-assessed disease activity.
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale
  Week 1 Day 7: number analyzed (Participants) | 38 | 107 | 108 | 110 | 107 | 47 | 47
  Week 1 Day 7 | -7.89 (13.16) | -10.68 (15.41) | -12.82 (17.03) | -5.85 (15.44) | -14.23 (16.13) | -9.57 (17.10) | -7.66 (18.33)
  Week 2 Day 14: number analyzed (Participants) | 39 | 106 | 109 | 110 | 109 | 48 | 48
  Week 2 Day 14 | -11.10 (15.65) | -15.86 (16.77) | -18.30 (19.04) | -9.01 (18.07) | -21.33 (19.61) | -14.23 (18.50) | -9.85 (17.55)
  Week 4 Day 28: number analyzed (Participants) | 38 | 104 | 106 | 108 | 108 | 47 | 48
  Week 4 Day 28 | -16.89 (19.06) | -22.02 (18.61) | -20.92 (17.71) | -14.01 (21.03) | -28.81 (19.34) | -17.70 (20.49) | -12.73 (20.42)
  Week 8 Day 56: number analyzed (Participants) | 37 | 101 | 103 | 102 | 108 | 47 | 44
  Week 8 Day 56 | -24.59 (15.06) | -28.52 (21.11) | -29.67 (20.01) | -20.87 (23.85) | -36.16 (21.82) | -22.40 (20.43) | -9.91 (19.67)
  Week 12 Day 84: number analyzed (Participants) | 37 | 98 | 96 | 102 | 107 | 47 | 45
  Week 12 Day 84 | -26.81 (16.20) | -32.43 (19.24) | -34.48 (19.49) | -23.19 (23.39) | -37.18 (21.02) | -30.82 (21.95) | -18.44 (21.86)

26. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) Levels
Description: C-reactive protein is a biological marker of inflammation and is measured in nanograms per milliliter (ng/mL)
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (ng/mL) nanograms per milliliter
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
(ng/mL) nanograms per milliliter
  Week 1 Day 7: number analyzed (Participants) | 37 | 106 | 107 | 109 | 107 | 47 | 46
  Week 1 Day 7 | 0.14 (2.09) | 0.30 (2.58) | 0.22 (2.49) | 0.01 (1.29) | -1.21 (2.37) | -0.12 (2.60) | -0.10 (1.76)
  Week 2 Day 14: number analyzed (Participants) | 38 | 106 | 108 | 110 | 109 | 48 | 47
  Week 2 Day 14 | 0.27 (1.78) | -0.10 (1.92) | -0.21 (2.29) | -0.12 (1.53) | -0.93 (2.70) | -0.20 (2.38) | -0.25 (2.60)
  Week 4 Day 28: number analyzed (Participants) | 37 | 103 | 105 | 105 | 109 | 47 | 48
  Week 4 Day 28 | 0.15 (2.45) | -0.25 (2.55) | -0.44 (2.30) | 0.14 (2.00) | -1.11 (2.17) | -0.30 (2.58) | -0.24 (2.80)
  Week 8 Day 56: number analyzed (Participants) | 36 | 100 | 103 | 100 | 106 | 47 | 45
  Week 8 Day 56 | -0.49 (1.66) | -0.52 (1.83) | -0.89 (3.16) | -0.39 (1.64) | -1.14 (2.39) | -1.19 (2.18) | -0.26 (2.55)
  Week 12 Day 84: number analyzed (Participants) | 37 | 97 | 97 | 102 | 106 | 47 | 44
  Week 12 Day 84 | -0.59 (1.43) | -0.77 (1.89) | -1.30 (2.88) | -0.45 (1.71) | -1.03 (2.01) | -1.55 (2.35) | -0.56 (2.75)

27. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: The Stanford Health Assessment Questionnaire disability index is a patient-reported outcome used to assess difficulty in performing activities of daily living. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities.
  To respond to each question, a four-level response with higher scores showing larger functional limitations, was chosen. Scoring is as follows with respect to performance of participant's everyday activities: 0 (equals)=without difficulties; 1= with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all. The composite HAQ-DI score is the mean of the eight domain scores and the score ranges from 0 (no functional impairment) to 3 (maximum functional impairment). A negative change from baseline indicates improvement.
Time Frame: Days 7, 14, 28, 56, and 84
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
Number analyzed (Participants) | 40 | 109 | 110 | 110 | 111 | 48 | 50
Score on a scale
  Week 1 Day 7: number analyzed (Participants) | 37 | 99 | 100 | 99 | 104 | 44 | 45
  Week 1 Day 7 | -0.20 (0.37) | -0.15 (0.35) | -0.22 (0.48) | -0.10 (0.38) | -0.26 (0.42) | -0.19 (0.36) | -0.14 (0.46)
  Week 2 Day 14: number analyzed (Participants) | 37 | 99 | 105 | 102 | 108 | 45 | 47
  Week 2 Day 14 | -0.24 (0.39) | -0.23 (0.46) | -0.28 (0.50) | -0.17 (0.45) | -0.35 (0.47) | -0.23 (0.45) | -0.13 (0.49)
  Week 4 Day 28: number analyzed (Participants) | 36 | 99 | 103 | 100 | 106 | 44 | 46
  Week 4 Day 28 | -0.34 (0.47) | -0.32 (0.48) | -0.40 (0.50) | -0.19 (0.56) | -0.50 (0.50) | -0.23 (0.42) | -0.17 (0.44)
  Week 8 Day 56: number analyzed (Participants) | 36 | 98 | 101 | 96 | 106 | 44 | 44
  Week 8 Day 56 | -0.49 (0.47) | -0.44 (0.56) | -0.56 (0.55) | -0.40 (0.64) | -0.60 (0.55) | -0.45 (0.50) | -0.23 (0.55)
  Week 12 Day 84: number analyzed (Participants) | 35 | 97 | 100 | 95 | 107 | 44 | 43
  Week 12 Day 84 | -0.51 (0.57) | -0.57 (0.57) | -0.65 (0.60) | -0.35 (0.68) | -0.65 (0.61) | -0.53 (0.61) | -0.30 (0.62)

28. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 to Time 24 of GDC-0853 at Steady State (AUC0-24,ss)
Description: The Pharmacokinetics (PK) evaluation may include, but will not be limited to, plasma GDC-0853 concentrations and population PK model estimated PK exposures (area under the plasma concentration-time curve [AUC]. AUC was measured in Nanograms(ng) per millilitre(mL)*hour (hr)
Time Frame: Pre-dose (0 hours) up to 10 hours post-dose on Day 28
Population: Intent-to-Treat (ITT) All randomized participants who received any part of an infusion of study medication were included in the ITT analysis. Number of participants for whom data were collected is indicated for each time point. Data were presented only for arms in which GDC-0853 was administered.
Measure: Mean (Standard Deviation); unit: Ng/mL*(hr)
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 2: GDC-0853 High Dose
Number analyzed (Participants) | 39 | 106 | 108 | 48
Ng/mL*(hr) | 1170 (1600) | 2910 (3180) | 9380 (4860) | 9890 (5480)

29. Secondary Outcome: Maximum Observed Plasma Concentration of GDC-0853 at Steady State (Cmax,ss)
Description: Cmax is the maximum (peak) plasma concentration over the dosing interval at steady state (ss)
Time Frame: Pre-dose (0 hours) up to 10 hours post-dose on Day 28
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Nanogram per Milliliter (ng/mL)
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 2: GDC-0853 High Dose
Number analyzed (Participants) | 39 | 106 | 108 | 48
Nanogram per Milliliter (ng/mL) | 110 (116) | 280 (223) | 591 (282) | 621 (302)

30. Secondary Outcome: Minimum Observed Plasma Concentration of GDC-0853 at Steady State (Cmin,ss)
Description: Cmin is the minimum concentration over the dosing interval at steady state (ss)
Time Frame: Pre-dose (0 hours) up to 10 hours post-dose on Day 28
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Nanogram per Milliliter (ng/mL)
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 2: GDC-0853 High Dose
Number analyzed (Participants) | 39 | 106 | 108 | 48
Nanogram per Milliliter (ng/mL) | 22.4 (41.0) | 54.7 (83.4) | 250 (146) | 263 (170)

ADVERSE EVENTS:
Time Frame: From randomization to end of study (approximately 22 months)
Arm/Group | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo | Cohort 1: GDC-0853 Placebo + Adalimumab | Cohort 2: GDC-0853 High Dose | Cohort 2: GDC-0853 Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/109 | 1/110 | 0/110 | 0/111 | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/40 | 1/109 | 3/110 | 1/110 | 2/111 | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 9/40 | 18/109 | 11/110 | 15/110 | 16/111 | 3/49 | 7/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo (N=40) | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo (N=109) | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo (N=110) | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo (N=110) | Cohort 1: GDC-0853 Placebo + Adalimumab (N=111) | Cohort 2: GDC-0853 High Dose (N=49) | Cohort 2: GDC-0853 Placebo (N=49)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
SMALL INTESTINAL DISORDERS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CELLULITS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS OBSTRUCTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: GDC-0853 Low Dose + Adalimumab Placebo (N=40) | Cohort 1: GDC-0853 Mid Dose + Adalimumab Placebo (N=109) | Cohort 1: GDC-0853 High Dose + Adalimumab Placebo (N=110) | Cohort 1: GDC-0853 Placebo + Adalimumab Placebo (N=110) | Cohort 1: GDC-0853 Placebo + Adalimumab (N=111) | Cohort 2: GDC-0853 High Dose (N=49) | Cohort 2: GDC-0853 Placebo (N=49)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 5 (5) | 3 (3) | 5 (6) | 1 (1) | 3 (4) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 6 (6) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (3) | 2 (3) | 0 (0) | 2 (2) | 8 (10) | 0 (0) | 3 (3)
ALANINE AMINOTRANFERASE INCREASED (Investigations) | 2 (3) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 4 (4) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 4 (5) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT02833350/Prot_SAP_001.pdf